

### **Clinical Trial Protocol**

Doc. No.: c02318676-08

2014-001687-36 EudraCT No.: **BI Trial No.:** 1311.13 **BI Investigational** BI 655066 **Product(s):** An open label extension trial assessing the safety and Title: Efficacy of BI 655066/ ABBV-066/risankizumab administered subcutaneously in patients with moderate to severe chronic plaque psoriasis. **Clinical Phase:** IIb **Trial Clinical** Monitor: Co-ordinating Investigator: **Status:** Final Protocol (Revised Protocol (based on global amendment 5) **Version and Date:** Version: 6.0 Date: 30-Jan-2018  Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

### **CLINICAL TRIAL PROTOCOL SYNOPSIS**

| Name of company: | | Tabulated Trial Day | |
|---|---|---|---|
| Boehringer Ingelheim | | Trial Protocol | |
| Name of finished produ | ict: | | |
| NA | | | |
| Name of active ingredic | ent: | | |
| BI 655066 | | | |
| Protocol date: 13 June 2014 | Trial number: 1311.13 | | Revision date: 30-Jan-2018 |
| Title of trial: | | on trial assessing the safety and eb administered subcutaneously in | |
| Co-ordinating<br>Investigator: | | poortusts. | |
| Trial site(s): | Multicenter, multination | onal | |
| Clinical phase: | IIb | | |
| <b>bjective(s):</b> Long term safety and efficacy of BI 655066/ ABBV-066/risankizumab dopen-label treatment in patients with moderate to severe chronic plaque psoriasis. | | | |
| Methodology: | Open label extension. | | |
| No. of patients: | 100 (estimated) | | |
| total entered: | 100 (estimated) | | |
| each treatment: | | ve 90 mg BI 655066/ ABBV-066<br>0 or 180 mg every 12 weeks depe | |
| Diagnosis : | Moderate to severe chi | ronic plaque psoriasis. | |
| Main criteria<br>for inclusion: | successfully completed preceding trial is defined a. Completion of t | e to severe chronic plaque psoria<br>d the preceding trial 1311.2. Suc<br>ted as either of the following:<br>he entire follow up period, thus to<br>e, defined as decrease in response | cessful completion of reaching EOS visit. |
| Test product(s): | BI 655066 | | |
| dose: | 90 mg every 12 weeks | , or 180 mg every 12 weeks | |
| mode of admin.: | Subcutaneous injection | n | |
| Comparator products: | NA | | |
| dose: | NA | | |

| Name of company: | | Tabulated | |
|---|---|---|---|
| Boehringer Ingelheim | | Trial Protocol | |
| Name of finished produ | ict: | | |
| NA | | | |
| Name of active ingredie | ent: | | |
| BI 655066 | | | |
| Protocol date:<br>13 June 2014 | Trial number: 1311.13 | | Revision date: 30-Jan-2018 |
| mode of admin.: | NA | | |
| Duration of treatment: | Approximately four years of administration to patient after receiving first BI 655066/ ABBV-066/risankizumab dose in either trial 1311.2 or trial 1311.13 | | |
| Criteria for efficacy: | | ASI <sub>90</sub> at week 48 in the Extended ASI score from baseline), is the | • • |
| Criteria for safety: Statistical methods: | safety. Safety analyses will for immune suppression a Analysis of laboratory of immune suppression Safety will also be ass tympanic body temper Additionally, time to a Kaplan Meier empirical | essed by evaluation of vital signs rature) and local tolerability. antibody development formation al survival curves. | early discontinuation, n hematologic measures s (BP, PR, RR, oral or will be examined using |
| Statistical methods: | will include a respond.<br>The analyses will be b<br>Kaplan Meier empirica | model; the analyses are descripti<br>er analysis, time to loss of respon-<br>assed on proportions of patients a<br>al survival curves to describe pat<br>as cumulative event rates at criti- | nse, and time to AESI.<br>achieving a response,<br>atterns of event |

30 January 2018

Boehringer Ingelheim BI Trial No.: 1311.13

Doc. No.: c02318676-08

Trial Protocol


# FLOW CHART - EXTENDED DOSING PERIOD

| Trial periods | | | | | Extended D | Extended Dosing Period | | | Extended FU period <sup>3</sup> |
|---|---|---|---|---|---|---|---|---|---|
| Visit | Extended<br>Visit 1 <sup>1, 2, 3</sup> | Extended<br>Visit 2 <sup>3</sup> | Extended<br>Visit 3 | Extended<br>Visit 4 | Extended<br>Visit 5 | Extended<br>Visit 6-<br>17 <sup>23</sup> | Extended<br>Visit 18<br>► | Extended<br>EOT <sup>4</sup> | Extended<br>EOS visit <sup>18,23</sup> |
| Day | - | 84 | 168 | 252 | 336 | 420-1344 | 1428<br><b>→</b> | X | Extended<br>EOT +84 |
| Week | 0 | 12 | 24 | 36 | 48 | 60-192 | 204 | X | Extended<br>EOT<br>+ 12 |
| Visit window (days) | | <i>1</i> ∓ | 77 | 7 | <del>1</del> 7 | 77 | <del>1</del> 7 | <del>1</del> 7 | -+4 |
| Informed Consent | x | | Ja - 15 | | | | | 8 | |
| Demographics <sup>20</sup> | х | | | | | | | | |
| Consent for vital status follow up <sup>20</sup> | 19 X | | | | | | | | |
| Med. history, smoking and alcohol use <sup>20</sup> | х | | | | | | | | |
| Psoriatic arthritis assessment /PASE <sup>5</sup> | × | | | | X | x S | | x | X |
| Weight, waist circum <sup>22</sup> | х | | | | X | $\mathbf{x}^{\mathbf{y}}$ | | × | x |
| Physical exam <sup>6,7</sup> | x <sub>C</sub> | LX | x <sub>C</sub> | X | xc | X I/C | $\mathbf{x}^{\mathbf{T}}$ | x <sub>C</sub> | X |
| Vital signs 8 | X | х | X | х | х | х | Х | Х | X |
| 12-Lead ECG9 | X | | × | | X | 6X | x | × | X |
| In/Ex eligibility <sup>20</sup> | Х | | | | | | | 95 37 | |
| Administer BI 6550663 | Х | X | X | Х | X | X | X | x <sub>10</sub> | |
| Adverse event 11 | X | X | X | X | X | X | X | Х | Х |
| Conc. Therapy | X | x | X | X | X | X | X | х | X |
| PASI <sup>3,21</sup> | PreD X | Y Card | $^{\rm PreD}_{\rm X}$ | $^{ m PreD}_{ m X}$ | $^{\rm PreD}_{\rm ~X}$ | $^{ m PreD}_{ m X}$ | PreD <sub>X</sub> | PreD <sub>X</sub> | х |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Boehringer Ingelheim BI Trial No.: 1311.13 Doc. No.: c02318676-08

Trial Protocol


| Trial periods | | | | | Extended D | Extended Dosing Period | | | Extended FU period <sup>3</sup> |
|---|---|---|---|---|---|---|---|---|---|
| Visit | Extended<br>Visit 1 <sup>1, 2, 3</sup> | Extended<br>Visit 2 <sup>3</sup> | Extended<br>Visit 3 | Extended<br>Visit 4 | Extended<br>Visit 5 | Extended<br>Visit 6-<br>17 <sup>23</sup> | Extended<br>Visit 18<br>► | Extended<br>EOT <sup>4</sup> | Extended<br>EOS visit <sup>18,23</sup> |
| Day | 1 | 84 | 168 | 252 | 336 | 420-1344 | 1428<br><b>→</b> | × | Extended<br>EOT +84 |
| Week | 0 | 12 | 24 | 36 | 48 | 60-192 | <del>2</del> 04 | × | Extended EOT + 12 |
| Visit window (days) | | 47 | ±7 | 77 | ±7 | <del>1</del> 7 | <b>1</b> 7 | ±7 | +7 |
| ${ m sPGA}^{21}$ | PreD X | PreD X | PreD X | PreD <sub>X</sub> | PreD X | PreD X | PreD <sub>X</sub> | PreD X | × |
| Pain VAS <sup>12,21</sup> | PreD X | PreD <sub>X</sub> | PreD X | PreD X | PreD X | PreD X | PreD X | PreD X | x |
| DLQI <sup>21</sup> | PreD X | PreD X | PreD X | PreD <sub>X</sub> | PreD <sub>X</sub> | PreD <sub>X</sub> | PreD X | PreD X | х |
| Local tolerability test | | PreD X | PreD <sub>X</sub> | PreD <sub>X</sub> | PreD <sub>X</sub> | $_{\rm X}^{\rm PreD}_{\rm X}$ | PreD <sub>X</sub> | PreD <sub>X</sub> | |
| Safety Lab 13, 14 | X | × | × | × | х | х | x | × | × |
| Serum pregnancy test<br>13, 15, 20, 24 | x | | | | | | | × | x <sup>24</sup> |
| TB screening 13, 20, 24 | х | | | | | | | × | x <sup>24</sup> |
| Urine Pregnancy test <sup>16</sup> | PreD X | PreD <sub>X</sub> | PreD <sub>X</sub> | PreD X | FreD X | $\Pr_{X}$ | PreD <sub>X</sub> | PreD <sub>X</sub> | × |
| PK <sup>17</sup> | PreD X | | PreD X | | FreD X | PreD I' | PreD <sub>X</sub> | PreD X | × |
| Anti-drug Ab (ADA)17 | PreD X | | PreD $_{ m X}$ | | PreD <sub>X</sub> | PreD $_{ m X}^{17}$ | PreD <sub>X</sub> | PreD <sub>X</sub> | X |
| Protein biomarker in plasma /serum <sup>17</sup> | PreD X | | PreD X | | PreD X | PreD $_{ m X}^{17}$ | PreD $_{ m X}$ | PreD X | x |
| M15-997 Open label extension study <sup>23</sup> | | | 2 | | | | | | X |
| Conclusion of patient<br>Participation | | | | | | | | | X |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Doc. No.: c02318676-08 BI Trial No.: 1311.13

# Footnotes:

- thereafter. If not performed as combined visits, informed consent must be signed before the roll-over visit due to lab sampling fasting at EV1 in trial 1311.13. Informed consent must not be Extended Visit 1 of this OLE study should preferably be performed in one visit combined with EOS visit in preceding trial 1311.2, or within an interim period of maximum 6 weeks signed before the 1311.2 date of last visit.
  - Assessments performed at EOS in the previous trial do not have to be repeated at EV1 in this trial, if performed as combined visits. If EV1 is performed as a separate visit to 1311.2 EOS, all EV1 assessments should be performed 7
- After the approval of this protocol amendment in each respective country, all patients will follow Flow Chart (Extended dosing period) and receive 90mg BI 655066 subcutaneously at their EVI. After 12 weeks, at EV2, the dose can be increased to 180 mg BI 655066 based on evaluation of the PASI90 achievement (see section 4.1.2 and 6.2.2). For ongoing patients under the previous protocol amendment, EV1 should be conducted at the following time points: ε.
- should not be conducted at the time point of Visit 2 under the previous protocol, patients with Visit 2 as their next scheduled visit should have their EV1 replacing their Visit 3 For ongoing patients still undergoing treatment or with <12 weeks since the EOT visit: Conduct EV1 at the time of the next scheduled treatment or follow up visit (note: EV1 For ongoing patients with  $\geq \! \! 12$  weeks since the EOT visit: Conduct EV1 as soon as possible
- taken at a regular study visit, the visit should be turned into an Extended EOT visit, i.e. an Extended EOT visit is to be performed instead of the scheduled visit. If the decision to discontinue For patients who prematurely discontinue the treatment period before study end (for any reason), an early Extended EOT visit is required. If the decision to discontinue study participation is Chart. This early Extended EOT visit will include the same procedures as the normal Extended EOT visit and the patient will subsequently enter a follow up period of 12 weeks, until a final study participation is taken in between study visits, an Extended EOT visit is to be scheduled at the earliest convenience and by the latest at the next upcoming visit according to the Flow 4.
- The Psoriatic Arthritis status assessment (PSOA: Psoriatic arthritis diagnosed, suspected, or not present) will be performed at roll-over visit only. Psoriatic arthritis screening and evaluation tool (PASE) to be completed by the patient if psoriatic arthritis is suspected or confirmed. To be repeated once per year until study end, i.e at EV1, EV5, EV10...
- "xC" is a complete physical examination including assessment of vital sign measurements, general appearance, and evaluation of all organ systems
- "xT" is a targeted physical examination including assessment of vital sign measurements, and evaluation of organ systems associated with AE(s) symptoms or laboratory abnormalities. Measured after 5 minutes of rest in the supine position. Measurements of vital signs should, if possible, always precede blood sampling. 9 7. 8
- Following dosing visits: Vital signs will be taken ~ 30 min predose, 5 minutes and 30 minutes after the dose is administered Extended visit 1: Vital signs will be taken  $\sim 30$  min predose, 5 minutes, and 1 hour after the dose is administered а.
  - Non-dosing visit (Extended EOS): Vital signs will be measured once per visit
- ECG to be performed after 5 minutes of rest in the supine position, at every 24 weeks, starting from EV1 (EV1, EV3, EV5...). Should, if possible, be performed prior to blood sampling. Not to be performed for patients who prematurely discontinue the treatment period
  - All new AEs as well as unresolved AE from the preceding trial 1311.2 should be followed up within this study.
    - Only for patients with psoriatic arthritis.
- For details of laboratory tests cf. Section 5.2.3, Table 5.2.3:1 and 5.2.3:2
- Patients must be fasting for at least 8 hours prior to collection of the safety laboratory samples.
  - Only applicable for women of childbearing potential.
- In women of childbearing potential urine pregnancy test has to be performed before each administration of study drug.
- For patients who prematurely discontinue the follow up period before study end (for any reason), an early Extended EOS visit is required. This early Extended EOS visit will include the same Blood samples for protein biomarker, PK and ADA will be drawn  $\sim 30$  min before the subcutaneous injection (PreD) at every 24 weeks, starting from EV1 (EV1, EV3, EV5...) procedures as the normal Extended EOS visit. 11. 12. 13. 14. 15. 16. 18.
  - Patients will be asked to give consent to be contacted (or for their primary care physician to be contacted) by the study team to obtain vital status information preferably at the time of study
- Only required at EV1 for patients who are having EV1 as their first 1311.13 visit
- All efficacy assessments should be performed pre-dose (PreD) 20. 21. 22.
- To be repeated once per year until study end (EV1, EV5, EV10...)

# © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. Proprietary confidential information.

30 January 2018  Trial Protocol Doc. No.: c02318676-08 **Boehringer Ingelheim** BI Trial No.: 1311.13

After 01-May-2018 and approval of this protocol amendment in each respective country patients who have completed the study without early treatment discontinuation will be offered to roll over to M15-997 open label extension (OLE) trial if they fulfill the in- and exclusion criteria for the M15-997 trial. Refer to section 6.2.3.

The next visit and also the last visit after 1st May and approval of this amendment will be Extended EOS visit. Termination of trial medication page should be completed in the eCRF and 23.

treatment completed registered in IRT.

24. For patients not prematurely discontinued.

Abbreviations: PreD = Prior to dose

© 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. Proprietary confidential information.

### **TABLE OF CONTENTS**

| TIT | LE P | PAGE | | 1 |
|---|---|---|---|---|
| CL | INIC | AL TR | IAL PROTOCOL SYNOPSIS | 2 |
| FLO | ow ( | CHART | T – EXTENDED DOSING PERIOD | 4 |
| | | | NTENTS | |
| AB | BRE | VIATI( | ONS | 12 |
| 1. | | | CTION | |
| | 1.1 | | CAL BACKGROUND | |
| | 1.2 | | PROFILE | |
| 2. | | | LE, OBJECTIVES, AND BENEFIT - RISK | |
| <b>4</b> • | | | ENT | 18 |
| | 2.1 | | ONALE FOR PERFORMING THE TRIAL | |
| | 2.2 | | L OBJECTIVES | |
| | 2.3 | | FIT - RISK ASSESSMENT | |
| 3. | DES | CRIP | ΓΙΟΝ OF DESIGN AND TRIAL POPULATION | 20 |
| | 3.1 | OVER | ALL TRIAL DESIGN AND PLAN | 20 |
| | | 3.1.1 | Administrative structure of the trial | |
| | | 3.1.2 | Data Monitoring Committee (DMC) | 23 |
| | 3.2 | DISCU | USSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF TROL GROUP(S) | 23 |
| | 3.3 | | CTION OF TRIAL POPULATION | |
| | 5.5 | 3.3.1 | Main diagnosis for study entry | |
| | | 3.3.2 | Inclusion criteria | |
| | | 3.3.3 | Exclusion criteria | 25 |
| | | 3.3.4 | Removal of patients from therapy or assessments | |
| | | | 3.3.4.1 Removal of individual patients | |
| | | | 3.3.4.2 Discontinuation of the trial by the sponsor | |
| 4. | TRE | EATMI | ENTS | 28 |
| | 4.1 | TREA | TMENTS TO BE ADMINISTERED | 28 |
| | | 4.1.1 | Identity of BI 655066 and comparator product(s) | |
| | | 4.1.2 | Method of assigning patients to treatment groups | |
| | | 4.1.3 | Selection of doses in the trial | |
| | | 4.1.4 | Drug assignment and administration of doses for each patient | |
| | | 4.1.5<br>4.1.6 | Blinding and procedures for unblinding<br>Packaging, labelling, and re-supply | |
| | | 4.1.0 | i ackaging, labening, and i e-supply | 50 |

| | 4.1.7 | Storage conditions | 30 |
|---|---|---|---|
| | 4.1.8 | Drug accountability | 30 |
| 4.2 | | | |
| | TREA | | 31 |
| | 4.2.1 | | |
| | 4.2.2 | | |
| | | · | |
| 4.3 | TREA | TMENT COMPLIANCE | 33 |
| VA] | RIABL | ES AND THEIR ASSESSMENT | 34 |
| 5.1 | EFFIC | CACY - PHARMACODYNAMICS | 34 |
| | 5.1.1 | Endpoints of efficacy | 34 |
| | | · · | |
| | 5.1.2 | • | |
| 5.2 | SAFE' | · | |
| | 5.2.2 | | |
| | 0,2,2 | | |
| | 5.2.3 | 1 | |
| | 5.2.4 | | |
| | 5.2.5 | | |
| 5.3 | ОТНЕ | v - 2 | |
| | | · · | |
| 5.4 | | | |
| 3.3 | | | 43 |
| | J.J.4 | * | |
| | | 5.5.2.2 Plasma sampling for assessment of anti-drug antibody | |
| | 4.3<br>VA<br>5.1 | 4.1.8 4.2 CONC TREA 4.2.1 4.2.2 4.3 TREA VARIABL 5.1 EFFIC 5.1.1 5.1.2 5.2.2 5.2.3 5.2.4 5.2.5 5.3 OTHE 5.3.1 5.3.2 5.3.3 5.4 APPR 5.5 DRUG | TREATMENT 4.2.1 Rescue medication, emergency procedures, and additional treatment(s) 4.2.2 Restrictions regarding concomitant treatment 4.2.2.1 Restrictions regarding vaccination 4.2.2.2 Restrictions on diet and life style 4.3 TREATMENT COMPLIANCE VARIABLES AND THEIR ASSESSMENT 5.1 Endpoints of efficacy. 5.1.1 Primary endpoint of efficacy 5.1.1.2 Secondary endpoints of efficacy 5.1.1.3 Further endpoints of efficacy 5.1.2 Assessment of efficacy. 5.2.1 Endpoint(s) of safety 5.2.1 Endpoint(s) of safety 5.2.1.3 Further endpoints of safety 5.2.1.4 Secondary endpoints of safety 5.2.2 Assessment of adverse events 5.2.2.1 Definitions of adverse events 5.2.2.2 Adverse event and serious adverse event reporting 5.2.3 Assessment of safety laboratory parameters 5.2.4 Electrocardiogram 5.2.5 Assessment of other safety parameters 5.3.1 Other endpoint(s) 5.3.2 Other assessment(s) 5.3.3 Pharmacogenomic evaluation. 5.4 APPROPRIATENESS OF MEASUREMENTS AND PHARMACOKINETICS 5.5.1 Plasma sampling for pharmacokinetic analysis |


| | | 5.5.3 | Analytical determinations | 44 |
|----|-----|--------|-----------------------------------------------|----|
| | 5.6 | BIOM | ARKER(S) | 44 |
| | | 5.6.1 | Endpoints based on biomarker(s) | |
| | | 5.6.2 | Methods of sample collection | |
| | | 5.6.3 | Analytical determinations | 45 |
| | 5.7 | PHAR | MACODYNAMICS | 45 |
| | | 5.7.1 | Pharmacodynamic endpoints | |
| | | 5.7.2 | Methods of sample collection | |
| | 5.8 | PHAR | MACOKINETIC - PHARMACODYNAMIC RELATIONSHIP | 46 |
| 6. | INV | ESTIG | SATIONAL PLAN | 47 |
| | 6.1 | VISIT | SCHEDULE | 47 |
| | 6.2 | DETA | ILS OF TRIAL PROCEDURES AT SELECTED VISITS | 47 |
| | | 6.2.1 | Screening and run-in period(s) | 47 |
| | | 6.2.2 | Treatment period(s) | |
| | | | 6.2.2.1 Rollover visit - Extended visit 1 | 47 |
| | | | 6.2.2.2 Extended Dosing Period | 48 |
| | | 6.2.3 | End of trial and Extended follow-up period | 49 |
| | | | 6.2.3.1 Vital status | 49 |
| 7. | STA | TISTI | CAL METHODS AND DETERMINATION OF | |
| | SAN | MPLE S | SIZE | 50 |
| | 7.1 | STATI | ISTICAL DESIGN - MODEL | 50 |
| | 7.2 | NULL | AND ALTERNATIVE HYPOTHESES | 50 |
| | 7.3 | PLAN | NED ANALYSES | 50 |
| | | 7.3.1 | Primary analyses | 50 |
| | | 7.3.2 | Secondary analyses | 50 |
| | | 7.3.3 | Safety analyses | 51 |
| | | 7.3.4 | Interim analyses | |
| | | 7.3.5 | Pharmacokinetic analyses | |
| | | 7.3.6 | Pharmacodynamic analyses | |
| | | 7.3.7 | Pharmacogenomic analyses | |
| | 7.4 | | LING OF MISSING DATA | |
| | 7.5 | | OMISATION | |
| | 7.6 | DETE | RMINATION OF SAMPLE SIZE | 52 |
| 8. | INF | ORME | D CONSENT, DATA PROTECTION, TRIAL | |
| | REC | CORDS | 5 | 53 |
| | 8.1 | | Y APPROVAL, PATIENT INFORMATION, AND INFORMED | |
| | 8.2 | | QUALITY ASSURANCE | |
| | 0.4 | DAIA | VUALITI ASSUNATICE | 33 |


| | 8.3 | RECORDS | 54 |
|---|---|---|---|
| | | 8.3.1 Source documents | 54 |
| | | 8.3.2 Direct access to source data and documents | 54 |
| | 8.4 | LISTEDNESS AND EXPEDITED REPORTING OF ADVERSE | |
| | | EVENTS | |
| | | 8.4.1 Listedness | 54 |
| | | 8.4.2 Expedited reporting to health authorities and IECs/IRBs | 54 |
| | 8.5 | STATEMENT OF CONFIDENTIALITY | 55 |
| | 8.6 | COMPLETION OF TRIAL | 55 |
| 9. | REF | TERENCES | 56 |
| | 9.1 | PUBLISHED REFERENCES | 56 |
| | 9.2 | UNPUBLISHED REFERENCES | |
| 10. | APP | PENDICES | 58 |
| | 10.1 | PASI SCORE DEFINITION AND INSTRUCTIONS | 58 |
| | 10.2 | STATIC PHYSICIAN'S GLOBAL ASSESSMENT (SPGA) OF THE | NPF |
| | | PSORIASIS SCORE (NPFPS) | |
| | 10.3 | PAIN VISUAL ANALOG SCALE (VAS) | 60 |
| | 10.4 | DERMATOLOGY LIFE QUALITY INDEX | |
| | 10.5 | PSORIATIC ARTHRITIS SCREENING AND EVALUATION TOO | L61 |
| | 10.6 | CLINICAL EVALUATION OF LIVER INJURY | 63 |
| | | 10.6.1 Introduction | 63 |
| | | 10.6.2 Procedures | 63 |
| | 10.7 | SEVERITY OF AE AS DESCRIBED IN THE RHEUMATOLOGY | |
| | | COMMON TOXICITY CRITERIA V. 2.0 | 65 |
| 11. | DES | CRIPTION OF GLOBAL AMENDMENT(S) | 90 |

### **ABBREVIATIONS**

ADA Anti-drug antibodies
ADL Activities of daily living

AE(s) Adverse event(s)

AESI Adverse event of special interest
ALT [U/L] Alanine transaminase (SGPT)
aPTT Partial Thromboplastin Time

AP/ALP Alkaline Phosphatase

AST [U/L] Aspartate transaminase (SGOT)

β Slope parameter associated with the power model used

to evaluate dose proportionality

BCG Bacille Calmette-Guérin vaccine

BI Boehringer Ingelheim

BP [mmHg] Blood pressure
BSA Body surface area
CA Competent Authority
Cf. Confer (compare)
CHF Congestive heart failure
CML Local clinical monitor

CRA Clinical research associate
CRO Clinical research organisation

CRF(s)
Case report form(s)
CRP
C-reactive protein
CTP
Clinical Trial Protocol
DILI
Drug-induced liver injury
DLQI
Dermatology Life Quality Index
DMC
Data monitoring committee

e.g. Example given ECG Electrocardiogram

eCRF(s) Electronic case report form(s)
EDTA Ethylendiaminetetraacetic acid

ELISA Enzyme-linked immunosorbent assay

EOS End of study
EOT End of treatment

Etc. Etcetera

EV Extended Visit

FDA Food and drug administration

FVC Forced vital capacity

g gram(s) (for description of mass);

gravity (description of centrifugation)

GCP Good clinical practice

30 January 2018

Doc. No.: c02318676-08 Trial Protocol 

Hb Haemoglobin

HbA1c Haemoglobin (glycated Hb of A1c subtype)

HCG Human chorionic gonadotropin

Hct Haematocrit

HDL High density lipoprotein

HIV Human immunodeficiency virus

i.e. Id est, that is

ICH International conference on harmonisation

IEC Independent ethics committee

IFN Interferon

IgG Immuneglobuline

IGRA Interferon gamma release assay

IL Interleukin

INR International normalised ratio IRB Institutional review board

IRT Interactive Response Technology

ISF Investigator site file

i.v. Intravenous

LLN Lower limit of normal mAb Monoclonal antibody

MACE Major Adverse Cardiovascular Events

MedDRA Medical dictionary for drug regulatory affairs

mg Milligrams ml Millilitre

mM Millimole/Millimolar

MRI Magnetic resonance imaging

NGAL Neutrophil gelatinase associated lipocalin

nM Nanomole/nanomolar

NPFPS National Psoriasis Foundation Psoriasis Score

OLE Open label extension OPU Operation Unit

OTC Over the counter medication

PASE Psoriatric Arthritis Screening and Evaluation Tool

PASI Psoriasis Area and Severity Index

PD Pharmacodynamic(s)
pH Power of hydrogen
PK Pharmacokinetic(s)
PMN Polymorphonuclear

PR [1/min] Pulse rate

PT Prothrombin time
PUVA Psoralen + UVA
RBC Red blood cell count

RCTC Rheumatology Common Toxicity Criteria

RDC Remote data capture

### Proprietary confidential information.

Trial Protocol 

REP Residual effect period RR Respiratory rate

SAE Serious adverse event

s.c. Subcutaneous

SOP Standard operating procedure

sPGA Static Physician Global Assessment

SUSARs Suspected unexpected serious adverse reactions

TB Tuberculosis

TCM Trial Clinical Monitor

Th Thelper (cell)
TMF Trial Master File
TNF Tumor necrosis factor
ULN Upper limit of normal

US United States
UVA Ultraviolet-A rays
UVB Ultraviolet-B rays
VAS Visual Analogue Scale
WBC White blood cells

### 1. INTRODUCTION

### 1.1 MEDICAL BACKGROUND

Psoriasis is a common skin disease characterized by raised, well-demarcated erythematous oval plaques with adherent silvery scales (<u>R11-1257</u>). It affects approximately 2% of the world population including 25 million people in North America and Europe making it the most prevalent immune mediated skin disease (<u>R08-1089</u>). It usually begins in late adolescence and early adulthood and then usually persists for life with remissions and relapses. The latter can be triggered by infections, medications and stress.

Disease severity can be characterized by body surface area (BSA) involvement with <5% being considered mild, 5-10% moderate and >10% severe (R11-1259). Disease status has been measured using the Psoriasis Area and Severity Index (PASI), a composite measure of erythema, induration, desquamation and BSA affected by psoriasis with a range of scores from 0 to 72 (R96-3541). The percentage of patients reaching PASI75, a 75% reduction in score from baseline to 12 or 16 weeks is traditionally used as a primary endpoint in psoriasis treatment trials.

Topical agents, including corticosteroids, are the mainstay for mild disease. Treatments for more advanced conditions can be classified into phototherapy, immunosuppressants, other systemic agents, and more recently, biologics (R11-1261).

Many of the agents may be used in combination or on a rotational basis to limit toxicity. Phototherapy may be used alone or with topical tar and dithranol products or with systemic and biologic agents. Although effective, the frequency and nature of this treatment reduces adherence. Adverse events (AEs) of phototoxicity, skin aging and concerns of development of skin cancers, also reduce acceptance of this therapy (R11-1261). Immunosuppressants, such as methotrexate or cyclosporine, are also effective for the management of moderate to severe psoriasis and relapses, but cumulative hepatotoxicity, bone marrow suppression and rarely pulmonary toxicity with methotrexate and nephrotoxicity with cyclosporine, requires careful monitoring and prevents the use of these agents long term.

Biologic agents such as tumor necrosis factor (TNF) blockers were first found efficacious in Crohn's disease, ulcerative colitis and rheumatoid arthritis prior to their use in psoriasis. Although not studied in head-to-head comparisons, different agents in this class have varying efficacy in psoriasis: infliximab and adalimumab are more efficacious especially in short term with PASI75 of 70-87% vs. etanercept (PASI75 of 50%) (R11-1261). These agents have been used for treating relapses and maintenance as well as the management of psoriatic arthritis, which occurs in approximately a third of all patients with psoriasis. However, TNF has myriad effects on immune function and TNF blockers have been associated with an increased risk of serious infections, in particular, tuberculosis and other opportunistic infections, cancers, including lymphomas, and demyelinating disorders.

BI 655066 is a humanized antagonistic monoclonal antibody (mAb) directed against the p19 subunit of the human cytokine interleukin-23 (IL-23). IL-23 plays a critical role in the

differentiation and function of Th17 cells, which have emerged as an important T-cell subpopulation involved in the pathogenesis of immune mediated disorders (R12-1008)

The therapeutic rationale for an IL-23 antagonist in inflammatory diseases such as psoriasis, Crohn's disease, and ankylosing spondylitis, is supported by several lines of evidence including mouse models, genome-wide association studies and histological findings in humans.

Although previous experience with selective IL-23 antagonists is limited, a mAb targeting the common p40 subunit of the IL-12 and IL-23 cytokines, ustekinumab (Stelara<sup>®</sup>), has been approved for the treatment of psoriasis, and a second (briakinumab) reached Phase III clinical trials before development was stopped. Both ustekinumab and briakinumab showed efficacy in the treatment of psoriasis.

The critical role of IL-12 in adaptive immunity raised concerns that mAbs directed against the IL-12 p40 subunit could increase the risk of infections or cancer, due to inhibition of IL-12-dependent immune surveillance mechanisms (<u>P06-11555</u>, <u>R11-1236</u>). Indeed, higher rates of these events were noted in pivotal Phase III randomised controlled trials of briakinumab (<u>R11-1529</u>, <u>R12-1010</u>), although not in trials of ustekinumab. However, complete IL-23 deficiency is not associated with a predisposition to mycobacterial infections (<u>R12-1011</u>) although it is associated with significant defects in humoral and delayed-type hypersensitivity responses in mice (<u>R11-1204</u>).

Observations of Major Adverse Cardiovascular Events (MACE) during the clinical development of both briakinumab and ustekinumab raised concerns that inhibition of either IL-12, IL-23, or both could pose cardiovascular safety risks (R11-4193). However, such a risk has not been confirmed among patients receiving ustekinumab for up to five years (R13-3518). No additional data has emerged to suggest a specific cardiovascular risk associated with inhibition of IL-23; nevertheless, particular attention will be given to cardiovascular AEs in clinical trials of BI 655066.

### 1.2 DRUG PROFILE

BI 655066 is a humanized monoclonal antibody (mAb) of the IgG1 subclass that is directed towards IL-23p19. The framework of the antibody has been engineered with two mutations in the Fc region to reduce Fc $\gamma$  receptor and complement binding. The C-terminal lysine of the heavy chain has also been deleted to reduce potential charge heterogeneity.

In Study 1311.1, a Phase I single rising dose trial in psoriasis patients, administration of BI 655066 either intravenously or subcutaneously appeared to be well tolerated. A total of 39 patients received a single dose of either BI 655066 i.v. (n=18), s.c. (n= 13), or placebo (n=8). All patients who received 0·01, 0·25, 3, or 5 mg/kg i.v., or 0·25 or 1 mg/kg s.c. doses of BI 655066 (n=27) achieved PASI<sub>75</sub> responses by Week 12 *vs.* 33% (1/3) and 67% (2/3) in 0·05 and 1 mg/kg i.v. dose groups, respectively *vs.* 13% (1/8) in the combined placebo group. PASI<sub>90</sub> rates by Week 12 were up to 100% (0·01 mg/kg i.v. group [3/3] and in both s.c. dose groups [13/13]) *vs.* 0% (0/8) in placebo group. Efficacy was well maintained at Week 24 and beyond. Treatment with BI 655066 resulted in significant changes in select psoriasis related

biomarkers in the skin and plasma through Week 12 and correlated with improvement in PASI scores. There were no clear relationships between the overall frequency of AEs and treatment; nor were there clear relationships between the occurrence of AEs in specific organ classes, individual AEs, their severity or relatedness, and treatment. Exposure increased in an approximately dose-proportional manner, with absolute bioavailability of 59%, providing a rationale for conducting further clinical studies of BI 655066 in patients with psoriasis. (M14-0004)

# 2. RATIONALE, OBJECTIVES, AND BENEFIT - RISK ASSESSMENT

### 2.1 RATIONALE FOR PERFORMING THE TRIAL

The phase I, single rising dose study (1311.1) has shown proof of concept and proof of efficacy for BI 655066 in patients with moderate to severe psoriasis.

The preceding phase II study (1311.2) will allow for the evaluation of the efficacy, safety, tolerability, pharmacokinetics and pharmacodynamics of three different dose regimens (18 mg, 90 mg and 180 mg) of BI 655066, as well as dose-finding of BI 655066 for further studies. In addition the 1311.2 trial will compare the efficacy of BI 655066 with Stelara<sup>®</sup>, an approved therapy for patients with moderate to severe psoriasis.

The data generated from this extension study is anticipated to provide additional safety data of up to approximately four years treatment in approximately 100 patients treated with BI 655066. Furthermore the study is being performed in order to allow extended access to a potential beneficial intervention, according to the principles laid down in the Declaration of Helsinki.

### 2.2 TRIAL OBJECTIVES

The overall purpose of this open label extension (OLE) trial is to assess long-term safety and efficacy (durability of response) of BI 655066 in patients with moderate to severe chronic plaque psoriasis. In addition, this study will provide an opportunity for subjects to have extended access to a proven active therapy for approximately four years administration.

The primary objective of the study is to investigate safety of BI 655066, in patients with moderate to severe chronic plaque psoriasis, receiving long-term treatment.

Additional objectives of this study are to further investigate long-term efficacy, tolerability, pharmacokinetics, pharmacodynamics and immunogenicity of BI 655066.

Study endpoints are listed in Section 5.

### 2.3 BENEFIT - RISK ASSESSMENT

Results of the Phase I study with BI 655066 (study 1311.1) suggest that a single injection intravenously or subcutaneously (i.v. or s.c.) of BI 655066 is associated with substantial and durable improvements in the cutaneous manifestations of psoriasis. At doses of 0.25 mg/kg intravenously and above, all active dose groups showed improvement in mean PASI scores of at least 75% from baseline by week 12, which lasted at least until week 24. Similar improvements were observed in both of the active BI 655066 subcutaneous dose groups (M14-0004).

Patients rolling over in this OLE will have completed the single blind 1311.2 study where 75% of all patients will have received BI 655066 at different dose levels. Based on the preliminary data from study 1311.1 described in <u>Section 1.2</u>, where good tolerability was

shown, and no drug related serious adverse events (SAE), patients are likely to benefit from participation in this study.

Risks of participating in this study include risks related to the trial specific procedures such as blood sampling, subcutaneous injection of study medication. Blood sampling and subcutaneous injections can cause local bruising, inflammation, and pain.

As with any immune modulating agent, BI 655066 has the potential to impair immune function resulting in a risk of infection. This will be addressed by clinical monitoring for AEs during the treatment and follow up periods. Interferon gamma (IFN- $\gamma$ ) release assay to *M. tuberculosis* will be obtained at the initial roll-over visit, in order to exclude or discontinue documented untreated patients with active or latent tuberculosis infection (TB). All patients will be re-tested at the Extended end of treatment visit in order to assess long-term impact of BI 655066 on *M. tuberculosis* exposure. Patients having current signs or symptoms of infection or history of serious infection will not be included in the study.

The role of IL-23 in tumour immunity is not well established at this time, but an increased risk of cancer from an IL-23 antagonist, though considered small, cannot be excluded.

Major adverse cardiovascular events (MACE), including myocardial infarction, cerebrovascular accident, and cardiovascular death, have been initially reported in association with the anti-IL-12/23 agents, ustekinumab and briakinumab, in patients with psoriasis. However, such a risk has not been confirmed among patients receiving ustekinumab for up to five years (R13-3518). The overall risk of MACE in the present study is considered to be low.

Local reactions to i.v. and s.c. administered biologic agents are uncommon, and are usually limited to redness, swelling or induration at the injection site. Manifestations of systemic hypersensitivity reactions include anaphylaxis, pruritus, hypotension, and respiratory distress. Both local and systemic hypersensitivity reactions are readily detectable, transient in nature, and manageable with standard medical treatment. No systemic hypersensitivity reactions have been reported with BI 655066 to date. Patients will be closely monitored 30 minutes to 1 hour after drug administration for signs of redness, swelling or hardness at the injection site or generalized itching, dizziness or difficulty breathing.

Although rare, a potential for drug-induced liver injury is under constant surveillance by sponsors and regulators. Therefore, this study requires timely detection, evaluation, and follow-up of laboratory alterations of selected liver laboratory parameters to ensure patients' safety (cf. section 10.4).

The study has been designed, and will be conducted in such a manner as to limit these risks as much as possible. In order to mitigate any safety signals as early as possible, an independent Data Monitoring Committee (DMC) will oversee this study. Since all patients will receive active treatment at a dose of, or greater than the projected marketed dose, most patients will likely have a benefit from participating in this study. Therefore, the benefit-risk assessment is considered appropriate for a clinical trial of an experimental therapy at this stage of development.

### 3. DESCRIPTION OF DESIGN AND TRIAL POPULATION

### 3.1 OVERALL TRIAL DESIGN AND PLAN

This open label extension trial (OLE), investigates the additional safety and efficacy of the 90 mg dose of BI 655066. Approximately 100 patients who meet the entry criteria are planned for inclusion in this trial, rolling over from the preceding 1311.2 trial. The treatment will be open label.

The treatment period will be approximately four years of administration starting with first administration of BI 655066 in either trial 1311.2 or 1311.13, followed by a 12 week follow up period. After 01-May-2018 and approval of this protocol amendment in each respective country, the next study visit will be the Extended EOS visit and therewith the last visit in this study. Patients who have completed the study without early treatment discontinuation will be offered to roll over to M15-997 open label extension (OLE) trial if they fulfill the in- and exclusion criteria for the M15-997 trial. Refer to section 6.2.3.

Patients rolling over from the preceding trial 1311.2 will have to complete the treatment period in that trial, or complete the entire trial including the follow up period, reaching end of study. If, during the follow up period of the preceding trial (at any visit from week 24 and onwards in trial 1311.2) loss of response is detected, the patient can roll over in this extension trial. For this, loss of response is defined as  $< PASI_{50}$ .

Extended visit 1 of this trial should preferably be performed as a combined visit the same day as End of Study visit of 1311.2, or within an interim period of maximum 6 weeks thereafter.

### 1311.2



Figure 3.1:1 Guideline for roll over of patients from 1311.2 to OLE study 1311.13

1

After the approval of this protocol amendment in each respective country, all patients will follow Flow Chart (Extended Dosing Period) and receive 90mg BI 655066 subcutaneously at their Extended visit 1 (EV1). From EV1 onwards, BI655066 will be administered subcutaneously every 12 weeks during the trial. At EV2, if there is a lack of response, defined as <PASI90, the dose should be increased to 180mg for the remainder of the trial (see Fig 3.1.2).

For ongoing patients under the previous protocol amendment (Pre-Extended Dosing Period, see Fig 3.1.3), EV1 should be conducted at the following time points:

- 1. For ongoing patients with ≥12 weeks since the EOT visit: Conduct EV1 as soon as possible
- 2. For ongoing patients still undergoing treatment or with <12 weeks since the EOT visit: Conduct EV1 at the time of the next scheduled treatment or follow up visit (note: EV1 should not be conducted at the time point of Visit 2 under the previous protocol, patients with Visit 2 as their next scheduled visit should have their EV1 replacing their Visit 3 instead)



Figure 3.1:2 Guideline for assessment of dose adjustment

<sup>\*</sup> EV stands for extended visit

<sup>\*\*</sup> Week 0 is the first scheduled visit after amendment approval.

| Trial periods | | | 7 | Treatment pe | riod | | | | Follow | Up period | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 11 | 2 | 3 | Interim<br>Contact | 4 | 5 | EOT | FU1 | FU 2 | FU3 | EOS<br>visit |
| Day | 1 | 42 | 84 | 126,<br>210,<br>294,<br>etc | 168 | 252 | 336 | | EOT<br>+168 | EOT<br>+252 | EOT<br>+336 |
| Week | 0 | 6 | 12 | 18,30,<br>42,<br>etc | 24 | 36 | 48 | EOT<br>+12 | EOT<br>+24 | EOT<br>+36 | EOT<br>+48 |
| Visit window (days) | +7 | <u>+</u> 7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 | ±7 |

Figure 3.1:3 Visit schedule Pre-Extended Dosing Period

If there are any tolerability issues, as assessed by the investigator, the patient will be discontinued.

The plaque psoriasis will be evaluated by PASI score at each visit. The standard clinical endpoints of PASI50, PASI75, PASI90 and PASI100 will be assessed at each visit based on the baseline PASI from 1311.2.

The end of study is defined as the date the last subject completes the Extended End-of-study visit.

### 3.1.1 Administrative structure of the trial

The trial is sponsored by AbbVie in the US and Boehringer Ingelheim (BI) ex-US.

The trial is planned to be conducted at sites participating in the 1311.2 trial, i.e. it will be conducted at approximately 24 sites in 4 different countries.

Boehringer Ingelheim has appointed a Trial Clinical Monitor (TCM), responsible for coordinating the activities required in order to manage the trial in accordance with applicable regulations and internal standard operating procedures (SOPs), directing the clinical trial team in the preparation, conduct and reporting of the trial and ensuring appropriate training and information for Local Clinical Monitors (CML), Clinical Research Associates (CRAs) and investigators of participating countries.

Data management will be done by BI according to BI SOPs and the Statistical Evaluation will be done by AbbVie according to their SOPs. For these activities a Trial Data Manager and a Trial Statistician have been appointed. A list of responsible persons will be available in the Trial Master File (TMF).

The organisation of the trial in the participating countries will be performed by the respective local BI-organisation (Operation Unit (OPU)) or by a Contract Research Organisation (CRO) with which the responsibilities and tasks have been agreed and a written contract filed before initiation of the clinical trial. In each OPU participating in this study, a CML will be appointed responsible for coordinating the activities required, in order to manage the trial in accordance with applicable regulations and internal SOPs in the countries covered by the respective BI OPU.

A Co-ordinating Investigator has been nominated to coordinate investigators at different sites participating in this multicentre, multinational trial. Tasks and responsibilities for the Coordinating Investigator will be defined in a written contract filed before initiation of the trial.

Details of the trial supplies including responsible institutions are given in <u>Section 4</u> of this protocol.

The Investigator Site File (ISF) will be maintained at the sites as required by local regulation and BI-SOPs. A copy of the essential ISF documents will also be kept as an electronic TMF document according to BI SOPs.

A central laboratory service and an Interactive Response Technology (IRT) vendor will be used in this trial. Details will be provided in IRT Manual and Central Laboratory Manual, available in ISF.

Safety will be monitored by an independent Data Monitoring Committee (DMC).

### 3.1.2 Data Monitoring Committee (DMC)

The trial will include the review of data by an external, independent DMC, including an independent statistician. The purpose of the DMC is to ensure the welfare of subjects participating in this trial is maintained by monitoring the trial for possible, untoward harmful effects or inappropriate frequency of adverse events for this class of medication. The DMC will evaluate and analyse accrued, unblinded safety and efficacy data in order to recommend whether the trial should continue, be modified or stopped due to safety or lack of efficacy concerns. For details regarding DMC structure and scheduled meetings, please consult the DMC charter.

Sponsor will agree with the DMC a set of strictly defined stopping criteria for the study level, to be included into the DMC Charter.

The final DMC Charter will be available before study initiation.

# 3.2 DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUP(S)

Study 1311.13 is designed as an open label extension clinical trial, and is expected to generate additional safety information to support the registration submission. As noted in section 4.1.3 below, the intermediate dose (90 mg) from the 1311.2 study will be used, with the option of moving to a higher dose (180 mg) if inadequate clinical activity is noted. Our goal in this study is to obtain safety and efficacy data following long-term drug administration. As an open-label study, we realize that no powered or controlled analysis can be obtained. However, we will be able to evaluate initial tendencies and at the same time permit our early study participants an opportunity to maintain access to a therapy that initially has shown the potential to have significant clinical benefit.

### 3.3 SELECTION OF TRIAL POPULATION

Eligible patients from trial 1311.2 will be offered participation in this OLE trial. The check for patient eligibility will be based upon a successful completion (cf. Section 3.3.2) of the previous trial and on signing the Informed Consent for the OLE.

A 40 % dropout rate from preceding trial is expected, leaving approximately 100 patients to be entered in this trial.

A log of all patients included into the study (i.e. having given informed consent) will be maintained in the ISF at the investigational site.

### 3.3.1 Main diagnosis for study entry

Moderate to severe chronic plaque psoriasis.

### 3.3.2 Inclusion criteria

- 1. Patients with moderate to severe chronic plaque psoriasis, who have successfully completed the preceding trial, 1311.2. Successful completion of preceding trial is defined as either of the following:
  - a. Completion of the entire follow up period, thus reaching End-of-study (EOS) visit
  - b. Loss of response, defined as decrease in response to <PASI<sub>50</sub> at any time from week 24.
- Patient must give informed consent and sign an approved consent form prior to any study procedures in accordance with Good Clinical Practice (GCP) and local legislation
- 3. Applicable only for female patients:

Negative urine pregnancy dip stick test at the roll-over visit, and if available at roll-over visit, negative

Serum \(\beta\)-Human Chorionic Gonadotropin (\(\beta\)-HCG) test (cf. Section 3.3.4.1).

In addition:

Women of childbearing potential (not surgically sterilized and between menarche and

1 year postmenopausal), that, if sexually active agree to use one of the appropriate medically accepted methods of birth control in addition to the consistent and correct use of a condom from date of the roll-over visit until 12 weeks after last treatment in this trial. Medically accepted methods of contraception's are: ethinyl estradiol containing contraceptives, diaphragm with spermicide substance, and intra-uterine-device.

OR

Female patients which have vasectomized sexual partner(s) (vasectomy at least 1 year prior to enrolment).

OR

Surgically sterilized female patients with documentation of prior hysterectomy, tubal ligation or complete bilateral oophorectomy.

OR

Postmenopausal women with postmenopausal is defined as permanent cessation  $\geq 1$  year of previously occurring menses.

### 3.3.3 Exclusion criteria

- 1. Patients who experienced any drug related Serious Adverse Event in the preceding trial
- 2. Patients who have developed guttate, erythrodermic or pustular psoriasis or druginduced psoriasis (as diagnosed by the investigator), during the preceding trial 1311.2.
- 3. Evidence of current or previous clinically significant disease, medical condition other than psoriasis, or finding of the medical examination (including vital signs and (electrocardiography (ECG)), that in the opinion of the investigator, would compromise the safety of the patient or the quality of the data.
- 4. Known clinically important acute or chronic infections including hepatitis, HIV. In regards to Tuberculosis the following applies:
  - Signs or symptoms suggestive of current active or latent tuberculosis upon medical history, physical examination and/or a chest radiograph (both posterior-anterior and lateral views, taken within 3 months prior to the first administration of study drug and read by a qualified radiologist).
  - History of latent or active TB prior to screening, except for patients with documented completion of an adequate treatment regimen, at least 6 months prior to the first administration of study agent.
  - Positive QuantiFERON-TB Gold In-Tube test (IGRA) within 2 months prior to the roll-over visit (if available) (cf. Section 3.3.4.1), in which active tuberculosis has not been ruled out. This does not apply to patients with history of latent tuberculosis with documented completion of an adequate treatment regimen, at least 6 months prior to the first administration of study agent.
- 5. Patients who have developed malignancy, or suspicion of active malignant disease during the preceding trial 1311.2 (except treated cutaneous squamous cell or basal cell carcinoma or carcinoma in situ of the cervix that have been adequately treated).

- 6. Intake of restricted medications (cf. <u>Section 4.2.2.1</u>) or other drugs considered likely to interfere with the safe conduct of the study, as assessed by the investigator.
- 7. Alcohol or drug abuse within 3 months prior to the roll-over visit that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures in the opinion of the investigator.
- 8. Any clinically significant laboratory abnormalities based on the last available lab results received during the preceding trial (according to the investigator's medical assessment) (cf. Section 6.2.2.1).
- 9. Pre-menopausal woman who is pregnant or nursing

### Note:

As there might be other medical and social issues, not covered by the above criteria it is left to the discretion of the investigator to exclude patients based on clinical judgment, even if other eligibility criteria are satisfied.

### 3.3.4 Removal of patients from therapy or assessments

### 3.3.4.1 Removal of individual patients

An individual patient is to be withdrawn from the trial if:

- The patient withdraws consent, without the need to justify the decision.
- Clinically important acute or chronic infections including hepatitis, HIV and tuberculosis (including latent tuberculosis), or a positive interferon gamma release assay (IGRA) testing for tuberculosis (cf. <u>Table 5.2.3: 1</u>) according to test at the roll-over visit.
- The patient is no longer able to participate for other medical reasons (e.g. pregnancy, surgery, AEs or other diseases).

A patient can be withdrawn after discussion between sponsor and investigator if eligibility criteria are being violated or if the patient fails to comply with the protocol (e.g. non-attendance at study assessments). Note: Patients using restricted medications (cf. Section 4.2.2), will continue to be followed up to collect safety data but their efficacy and PD endpoints assessed after administration of restricted medications will not be considered for analysis.

If a patient withdraws from the study after informed consent, this will be documented and the reason for withdrawal will be recorded in the case report form (CRF). This data will be included in the trial database and will be reported. At the time of discontinuation a complete end of treatment (Extended EOT) evaluation should be performed according to <u>Flow Chart</u> and the patient will subsequently enter a follow up period of 12 weeks, until a final Extended EOS visit is performed. If the decision to discontinue study participation is taken in between study visits in the treatment period, an Extended EOT visit is to be scheduled at the earliest convenience and by the latest at the next upcoming visit according to <u>Flow Chart</u> and the information will be recorded in the CRFs.

If the decision to discontinue is taken in the 12 week follow up period, an early Extended EOS visit is to be scheduled at the earliest convenience. The procedures described at Extended EOS will be performed and the information will be recorded in the CRFs. The withdrawals will be discussed in the final report of the study.

If a patient becomes pregnant during the trial, the investigational product needs to be stopped. The patient will be followed up until birth or otherwise termination of the pregnancy. The data of the patient will be collected and reported in the clinical trial report until last patient last visit and any events thereafter will be reported in the BI 655066 safety database.

### 3.3.4.2 Discontinuation of the trial by the sponsor

AbbVie/ Boehringer Ingelheim reserves the right to discontinue the trial overall or at a particular trial site at any time for the following reasons:

- a. Emergence of any efficacy/safety information that could significantly affect continuation of the trial or any other administrative reasons.
- b. Violation of GCP, the clinical trial protocol (CTP), or the contract by a trial site or investigator, disturbing the appropriate conduct of the trial.

The investigator / the trial site will be reimbursed for reasonable expenses incurred in case of trial termination according to option a.

### 4. TREATMENTS

### 4.1 TREATMENTS TO BE ADMINISTERED

BI 655066 is supplied by Boehringer Ingelheim, and will be administered subcutaneously.

### 4.1.1 Identity of BI 655066 and comparator product(s)

The characteristics of the test product for s.c. administration are below.

| Substance: | BI 655066: Anti-human IL23p19 mAb |
|---|---|
| Pharmaceutical formulation: | |
| Chemical name: | Anti-human IL-23p19 mAb |
| Molecular weight: | Approximately 148 kDa |
| Source: | Boehringer Ingelheim Pharma GmbH & Co. KG |
| Unit strength: | 90 mg BI 655066 in a pre-filled syringe with 1 ml (concentration 90 mg/ml) |
| Posology | Multiple doses |
| Route of administration: | s.c. |

### 4.1.2 Method of assigning patients to treatment groups

Patients will receive a single dose of open label BI 655066 every 12 weeks. The initial dose for all patients moving into the open label extension study will be 90 mg.

If response is maintained, i.e. achievement of PASI<sub>90</sub> at Extended visit 2, 90 mg dosing will occur every 12 weeks until Extended EOT.

If there is a lack of response, defined as response below PASI<sub>90</sub> at Extended visit 2, the dose should be increased to 180 mg, and the 180 mg dosing will occur every 12 weeks until Extended EOT.

Detailed instructions for preparation of BI 655066 for administration of each dose will be given in the ISF.

### 4.1.3 Selection of doses in the trial

The treatment is derived from the treatment groups in the preceding phase II trial, where the dose selection is based on the completed phase I trial in which clinical improvement in patients with psoriasis was observed across a wide dose range (~18 mg -375 mg).

The choice of the "90 mg/dose" was based on several pieces of data obtained in the initial 1311.1 single-dose, dose-escalation study: an analysis of dose given (and the subsequent "area under the curve" exposure data) plotted against the clinical response based on the PASI

score noted that the stable effective dose was likely to be greater than 1.0 mg/kg (approximately 90 mg)

Subsequent to selection of the starting dose for 1311.13, an interim analysis of 1311.2 indicated that the 180 mg dose resulted in a numerically higher proportion of patients who achieved PASI90. Since the higher dose was not associated with a higher incidence of any specific adverse events, patients who do not achieve PASI90 on the 90 mg dose are eligible to receive the higher dose of 180 mg. This dose is also consistent with the objective of obtaining safety data on a dose equal to or greater than the proposed "to be marketed" dose of 150 mg, allowing us to obtain additional safety information appropriate for inclusion in future discussion with health authorities.

### 4.1.4 Drug assignment and administration of doses for each patient

The study drug will be administered by the physician investigator or by authorised study personnel (e.g. study nurse). The study drug will be administered as a subcutaneous injection in the abdomen, thighs, gluteal regions, or upper arms. Injections being given in the same area should be at least 2 cm apart and should not be close to a vein. The injection site should avoid sites of psoriasis involvement as well as sites where the skin is tender, bruised, erythematous, or indurated, and should be alternated to other areas for subsequent doses.

Further information regarding technique of injection and injection materials (syringes, needles) will be provided in the ISF. For 180 mg doses, two syringes of 1 ml BI 655066, each of 90 mg, will be allocated and injected. Dilution of the study medication is not allowed and no dose modification, apart from the protocol specified doses, is permitted.

Administration of biologic agents involves the risk of local (injection site) or systemic hypersensitivity reactions. Therefore the patients should be closely monitored for signs and symptoms of hypersensitivity reactions for approximately 1 hour after the first dose administered, and 30 minutes following all other doses of study drug. Study personnel should observe the injection site for signs of redness, swelling or hardness. They should also ask subjects about itching, dizziness or shortness of breath. Patients should be advised that if they experience redness, swelling or other changes at the injection site, they should notify site personnel. They should further be advised that if they experience itching all over or a feeling of being swollen, dizzy or short of breath, they should notify site personnel or their own healthcare provider immediately.

Vital signs will be taken pre-dose, 5 minutes, and 1 hour (at roll-over visit) or 30 minutes (at following visits) after the dose is administered (cf. <u>Flow Chart</u>). Hypersensitivity reactions should be treated according to medical standards. Pre-medications for further injections might be considered and will be agreed on between investigator and BI clinical monitor.

### 4.1.5 Blinding and procedures for unblinding

Not applicable.

In this open-label trial, treatment allocation will not be concealed throughout the study. The CRF will contain information on treatment.

### 4.1.6 Packaging, labelling, and re-supply

BI 655066 supplies will be provided by Boehringer Ingelheim (cf. Section 4.1.1 for more details regarding the supplies). Pre-filled syringes of study medication will be provided in individual boxes identified with the trial number, batch and medication number. Supply of study medication will be managed by the IRT.

For details of packaging and the description of the label, refer to the ISF.

### 4.1.7 Storage conditions

The trial medication must be stored securely, e.g. in a locked refrigerator or at a pharmacy, in their original packaging. It may only be dispensed to trial patients according to the clinical trial protocol, by authorised personnel as documented in "Trial Staff List".

Drug supplies should be stored as indicated on the country specific booklet page. A temperature log must be maintained. If the storage conditions are found to be outside the specified range, immediately contact the local clinical monitor as provided in the lists of contacts.

Further details are provided in the Investigator's Brochure and on the country specific labels of which a sample will be maintained in the ISF.

### 4.1.8 Drug accountability

The investigator/ pharmacist/ investigational drug storage manager will receive the investigational drugs delivered by the sponsor when the following requirements are fulfilled:

- approval of the study protocol by the Institutional Review Board (IRB) / ethics committee,
- availability of a signed and dated clinical trial contract between the sponsor and the Head of Trial Centre,
- approval/notification of the regulatory authority, e.g. competent authority,
- availability of the curriculum vitae of the principal investigator,
- availability of a signed and dated clinical trial protocol or immediately imminent signing of the clinical trial protocol,
- availability of the proof of a medical licence for the principal investigator,
- availability of the Form 1572 (only applicable for (United States (US)).

The investigator/ pharmacist/ investigational drug storage manager must maintain records of the product's delivery to the trial site, the inventory at the site, the use by each patient, and the return to the sponsor or alternative disposition of unused product(s), on the respective forms in the ISF.

These records will include dates, quantities, batch/serial numbers, expiry ('use by') dates, and the unique code numbers assigned to the investigational product(s) and trial patients. The

investigator / pharmacist / investigational drug storage manager will maintain records that document adequately that the patients were provided the doses specified by the CTP and reconcile all investigational product(s) received from the sponsor. At the time of return to the sponsor or designee, the investigator / pharmacist / investigational drug storage manager must verify that all unused or partially used drug supplies have been returned and that no remaining supplies are in the investigator's possession. Account must be given for any discrepancies.

## 4.2 CONCOMITANT THERAPY, RESTRICTIONS, AND RESCUE TREATMENT

### 4.2.1 Rescue medication, emergency procedures, and additional treatment(s)

In principle, any additional concomitant therapy considered necessary for the patient's welfare may be given at the discretion of the investigator. Stable doses of concomitant therapies for chronic conditions, for which neither the condition nor the treatment are judged to exclude the patient from participation (cf. Section 3.3.3), are permissible. However, all concomitant medications being taken by eligible patients must be carefully evaluated, and questions on the use of concomitant medications should be discussed with the BI clinical monitor.

In the event that a patient experiences an intolerable increase of psoriasis during the course of the trial, topical steroids of US class 6 (mild, such as desonide) or US class 7 (least potent, such as hydrocortisone) will be permitted for use limited to the face, axilla, and/or genitalia. Details of the drug used and the reason must be recorded in the electronic case report forms (eCRF). These topical medications should not be used within approximately 24 hours prior to visits requiring the PASI.

Investigational products are not allowed during the course of the trial.

In case of adverse events in need of treatment, symptomatic therapy according to the judgment of the investigator will be permitted. All concomitant and/or rescue therapies will be recorded on the appropriate pages of the eCRF.

There are no special emergency procedures to be followed.

Patients with a positive IGRA testing (Tb screening) at the roll-over visit should be followed-up according to local guidelines.

### 4.2.2 Restrictions

### 4.2.2.1 Restrictions regarding concomitant treatment

The medications (or classes of medication) listed in <u>Table 4.2.2.1:1</u> must not be taken for the specified times before the roll-over l visit and for the whole duration of the study including the Extended Follow-up Period.

Table 4.2.2.1: 1 Restricted medications

| Investigational products not otherwise | Throughout the duration of preceding trial |
|---|---|
| described below (except 1311.2 study drug) | 1311.2, and for the whole duration of this |
| | trial, including any interim period between |
| | the trials and the Extended Follow-up Period. |
| Any biological agents, including but not | Throughout the duration of preceding trial |
| limited to infliximab, etanercept, | 1311.2, and for the whole duration of this |
| adalimumab | trial, including any interim period between |
| | the trials and the Extended Follow-up Period |
| Oral or injectable psoriasis medications (not | Throughout the duration of preceding trial |
| biologicals) including but not limited to | 1311.2, and for the whole duration of this |
| retinoids, methotrexate, cyclosporine, | trial, including any interim period between |
| fumarates, or any other drugs known to | the trials and the Extended Follow-up Period |
| possibly benefit psoriasis. | |
| Systemic corticosteroids in any dosage form. | |
| Any drug known to interfere with or to | |
| aggravate psoriasis including but not limited | |
| to lithium and interferons, or | |
| Phototherapy (UVB, PUVA, UVA). | |
| Steroids, retinoids, vitamin D analogs, | Throughout the duration of preceding trial |
| vitamin A analogs and anthralin in any | 1311.2, and for the whole duration of this |
| formulation (i.v., s.c., topicals, oral). | trial, including any interim period between |
| | the trials and the Extended Follow-up Period. |
| | (for exceptions cf. <u>Section 4.2.1</u> ) |

### 4.2.2.2 Restrictions regarding vaccination

Live vaccinations during the study are not allowed. Bacille Calmette-Guérin vaccines (BCG) are not allowed throughout the duration of preceding trial 1311.2, and for the whole duration of this trial, including any interim period between the trials. It is recommended that patients are advised not to take any live vaccines or BCG vaccines for up to 1 year after the last administration of study drug.

### 4.2.2.3 Restrictions on diet and life style

Patients must be fasted for at least 8 hours prior to collection of the safety laboratory samples, starting from the initial roll-over visit.

Patients should refrain from excessive physical activity at least 24 hours prior to study visits, during the course of the study (competitive sport etc.).

Use of tanning beds is not allowed during the course of the study.

### 4.3 TREATMENT COMPLIANCE

Dose administration compliance will be assured by administration of all study medication under supervision of the investigating physician or a designee at the research site. The measured plasma concentrations will provide additional information about compliance.

### 5. VARIABLES AND THEIR ASSESSMENT

### 5.1 EFFICACY - PHARMACODYNAMICS

### 5.1.1 Endpoints of efficacy

### 5.1.1.1 Primary endpoint of efficacy

The primary efficacy endpoint is achievement of a  $\geq$  90% reduction in PASI score from baseline (i.e., achieving PASI<sub>90</sub>) at week 48 in the Extended dosing period. Baseline PASI for this study is defined as the baseline PASI for the 1311.2 study.

### 5.1.1.2 Secondary endpoints of efficacy

The following secondary endpoints will all be evaluated at week 48in the Extended dosing period:

- achievement of PASI<sub>50</sub>
- achievement of PASI<sub>75</sub>
- achievement of PASI<sub>100</sub>
- achievement of sPGA of clear or almost clear

### 5.1.1.3 Further endpoints of efficacy

Additional efficacy analyses will include, but are not limited to, the following:

- achievement of PASI<sub>50</sub> at all Extended dosing period visits where PASI is collected
- achievement of PASI<sub>75</sub> at all Extended dosing period visits where PASI is collected
- achievement of PASI<sub>90</sub> at all Extended dosing period visits where PASI is collected
- achievement of PASI<sub>100</sub> at all Extended dosing period visits where PASI is collected
- achievement of sPGA of clear or almost clear at all visits where sPGA is collected
- time to loss of PASI<sub>50</sub>, which is a time to failure endpoint. This will be repeated using PASI<sub>75</sub>, PASI<sub>90</sub>, and PASI<sub>100</sub> as the endpoint.
- sPGA will be evaluated in terms of time to loss of response which is defined as a score exceeding 1, and will be evaluated as a time to failure endpoint
- change from baseline in Pain-VAS (in subgroup of patients with psoriatic arthritis only where baseline VAS is from 1311.2)
- mean DLQI scores at all Extended dosing period visits where PASI is collected

### 5.1.2 Assessment of efficacy

The PASI measures the severity of a patient's psoriasis and the percent of the patient's skin that is affected. See <u>Section 10.1</u> for a detailed description of the PASI.

The Static Physician Global Assessment (sPGA) is a 6 point scale used by physicians to describe the severity of a patient's psoriasis. See <u>Section 10.2</u> for a detailed description of the sPGA.

The Pain-VAS is a Visual Analogue Scale used to assess a patient's psoriatic arthritis. See Section 10.3 for a detailed description of the Pain-VAS.

Immunogenicity testing (Anti-Drug Antibodies (ADA)) will be performed at the visits specified in the Flow Chart in order to detect the emergence of antibodies.

The Dermatology Life Quality Index (DLQI) is a questionnaire that determines a patient's quality of life. See Section 10.4 for a detailed description of the DLQI.

### 5.2 SAFETY

### 5.2.1 Endpoint(s) of safety

### 5.2.1.1 Primary endpoints of safety

The primary endpoints of safety are as follows:

- the occurrence of AEs
- the occurrence of drug related AEs
- the occurrence of SAEs

### 5.2.1.2 Secondary endpoints of safety

Not applicable as there are no secondary endpoints of safety.

### 5.2.1.3 Further endpoints of safety

Safety and tolerability will be assessed in a descriptive way based on:

- Changes in vital signs and physical examination
- Adverse events (AEs)
- The occurrence of Adverse events of special interest (AESIs)
- Discontinuation of therapy due to AEs, SAE
- Changes in safety laboratory analysis

Immunogenicity testing (ADA) will be performed at the visits specified in Flow Chart in order to detect the emergence of antibodies. Immunogenicity will be evaluated in terms of time to antibody emergence starting from the time of first exposure to BI 655066 in either 1311.2 or 1311.13.

### 5.2.2 Assessment of adverse events

### 5.2.2.1 Definitions of adverse events

### Adverse event

An adverse event (AE) is defined as any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a patient in a clinical investigation who received a

### Proprietary confidential information.

pharmaceutical product. The event does not necessarily have to have a causal relationship with this treatment.

### Serious adverse event

A serious adverse event (SAE) is defined as any AE which results in death, is immediately life-threatening, results in persistent or significant disability / incapacity, requires or prolongs patient hospitalisation, is a congenital anomaly / birth defect, or is to be deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgement which may jeopardise the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions.

### Intensity of adverse event

The intensity grading of AEs will be performed according to Rheumatology Common Toxicity Criteria (RCTC) Version 2.0 developed by Outcome Measures in Rheumatology (OMERACT) (R13-3515). Cf. Appendix 10.7 and ISF for intensity/severity classification.

### Causal relationship of adverse event

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history. Assessment of causal relationship should be recorded in the case report forms.

Yes: There is a reasonable causal relationship between the investigational product administered and the AE.

No: There is no reasonable causal relationship between the investigational product administered and the AE.

### Worsening of the underlying disease or other pre-existing conditions

Worsening of the underlying disease or of other pre-existing conditions will be recorded as an (S)AE in the (e)CRF.

### Changes in vital signs, ECG, physical examination, and laboratory test results

Changes in vital signs, ECG, physical examination and laboratory test results will be recorded as an (S)AE in the (e) CRF, if they are judged clinically relevant by the investigator.

### Adverse Events of Special Interest (AESI)

The following are considered as Adverse events of Special Interest (AESI):

Hepatic injury defined by the following alterations of liver parameters (for patients with normal liver function at baseline): an elevation of AST and/or ALT  $\geq$ 3 fold upper limit of normal (ULN) combined with an elevation of total bilirubin  $\geq$ 2 fold ULN measured in the
same blood draw sample.

Patients showing these lab abnormalities need to be followed up according to section 10.6 of this clinical trial protocol and the "Drug induced liver injury (DILI) checklist" provided in ISF.

Major adverse cardiovascular events (MACE).
 Including, but not limited to the following preferred terms: Atherosclerosis, Coronary artery disease, Myocardial infarction, Angina Pectoris, Transient ischemic attack, Cerebrovascular accident (including Stroke), Cardiac failure congestive, Peripheral arterial occlusive disease.

ASEIs are to be reported in an expedited manner similar to Serious Adverse Events, even if they do not meet any of the seriousness criteria – for details please see section 5.2.2.2.

#### 5.2.2.2 Adverse event and serious adverse event reporting

All adverse events, serious and non-serious, occurring during the course of the clinical trial (i.e., from signing the informed consent onwards through the Residual Effect Period (REP) /Extended follow-up period) will be collected, documented and reported to the sponsor by the investigator on the appropriate CRF(s) / eCRFs / SAE reporting forms. Reporting will be done according to the specific definitions and instructions detailed in the 'Adverse Event Reporting' section of the Investigator Site File.

Reporting of Adverse Events in Remote Data Capture system (RDC):

AEs that are ongoing at the end of the previous trial (1311.2) will have to be re-entered, and any adverse events that have started between the two trials (in the event that the 6 weeks time-window is used), will also be entered into the 1311.13 RDC system.

Reporting of Adverse Events on the SAE form:

Specific instructions for the SAE reporting process concerning SAE forms in previous and roll-over studies will be provided in the ISF.

The REP for BI 655066 is 12 weeks. Therefore, all events reported within 12 weeks of the last trial medication will be considered on treatment. All adverse events will be reported up until the last per protocol visit (Extended EOS visit), which is 84 (+7 days) days after the last dose of trial medication.

The investigator does not need to actively monitor patients for AEs once the clinical trial has ended. However, if the investigator becomes aware of an SAE(s) that occurred after the patient has completed the clinical trial (including any protocol required REP and / or follow-up), it should be reported by the investigator to the sponsor if considered relevant by the investigator.

For each adverse event, the investigator will provide the onset date, end date, intensity, treatment required, outcome, seriousness, and action taken with the investigational drug. The

investigator will determine the relationship of the investigational drug to all AEs as defined in Section 5.2.2.1.

The investigator must report the following events using paper process SAE form via telephone/fax immediately (within 24 hours) to the sponsor: SAEs and non-serious AEs relevant to the SAE(s), and AESIs.

Boehringer Ingelheim has set up a list of AEs which are defined to be always serious. In order to support the investigator with the identification of these "always serious adverse events", if a non-serious AE is identified to be serious per Boehringer Ingelheim definition, a query will be raised. The investigator must verify the description and seriousness of the event. If the event description is correct, the item "serious" needs to be ticked and an SAE has to be reported in expedited fashion following the same procedure as above.

The list of these adverse events can be found via the RDC-system.

With receipt of any further information to these events, a follow-up SAE report has to be provided. SAEs and non-serious AEs must include a causal relationship assessment made by the investigator.

The SAE form is to be forwarded to the defined unique entry point identified for the BI OPU (country-specific contact details will be provided in the Investigator Site File) or by using the electronic submission process. This immediate report is required irrespective of whether the investigational product has been administered or not and irrespective of causal relationship. It also applies if new information to existing SAEs or AESIs becomes available.

# Pregnancy

In rare cases, pregnancy might occur in clinical trials. Once a female subject has been enrolled into the clinical trial, after having taken study medication, the investigator must report immediately any drug exposure during pregnancy to the sponsor. Drug exposure during pregnancy has to be reported immediately (within 24 hours or next business day whichever is shorter) to the defined unique entry point for SAE forms of the respective BI OPU (country-specific contact details will be provided in the Investigator Site File). The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up. In the absence of an (S)AE, only the Pregnancy Monitoring Form for Clinical Trials and not the SAE form is to be completed. The ISF will contain the Pregnancy Monitoring Form for Clinical Trials (Part A and Part B).

# 5.2.3 Assessment of safety laboratory parameters

The laboratory parameters that will be determined are listed in <u>Tables 5.2.3: 1</u> and <u>5.2.3: 2</u> at the time points provided in <u>Flow Chart</u>. The respective reference ranges will be provided in the ISF. The laboratory tests will be performed at a designated central laboratory, and if necessary by additional specialist laboratories.

Laboratory results of the patients will be available in real time to the respective investigator and to the clinical monitor of each country (central laboratory website), and selected

abnormal laboratory alerts will be sent automatically to the sites and to the sponsor in real time. PK, PD and biomarker data will not be available to the investigators or local clinical monitors, but only to the Trial Team (sponsor) and to the DMC.

Clinically relevant laboratory values will be commented on in the eCRF. A clinically relevant value may be either in- or outside the reference range. Clinically relevant abnormal laboratory test results must be repeated using an unscheduled visit lab kit and must be repeated until normalisation or stabilisation or until an alternative explanation has been found. Clinically relevant abnormal laboratory values will be also graded for intensity by using RCTC Version 2.0 criteria.

The tests listed in Table 5.2.3: 1 constitute laboratory tests and hormones (assessed in female patients only) that will be done only at the initial roll-over visit and at Extended EOT or Extended EOS after approval of amendment # 5 and start of the rollover of patients to the M15-997 study from 01-May-2018, i.e. these tests are only required at EV1 for patients that are having EV1 as their first 1311.13 visit. The results will not be included into the report. Samples will be archived and run as clinically necessary.

Table 5.2.3: 1 Exclusionary Testing

| Category | Test name |
|---|---|
| Tb screening | Interferon-gamma release assay (IGRA) |
| Serum pregnancy test (only female patients of childbearing potential) | Serum β-Human Chorionic Gonadotropin |

Table 5.2.3: 2 Safety laboratory tests

| Category | Test name |
|---|---|
| Haematology | Haematocrit (Hct) Haemoglobin (Hb) Red Blood Cell Count / Erythrocytes Reticulocyte Count White Blood Cells / Leucocytes Platelet Count / Thrombocytes |
| | HbA1c (Haemoglobin (glycated Hb of A1c subtype))<br>Roll-over and final visits only |

Table 5.2.3: 2 Safety laboratory tests (cont'd)

| Category | Test name |
|---|---|
| Diff Automatic | Neutrophils (relative and absolute count) Eosinophils (relative and absolute count) Basophils (relative and absolute count) Monocytes (relative and absolute count) Lymphocytes (relative and absolute count) |
| Diff Manual<br>(if Diff Automatic is abnormal) | Neutrophils, Bands (Stabs) Neutrophils, Polymorphonuclear (PMN) Eosinophils Basophils Monocytes Lymphocytes |
| Coagulation | Partial Thromboplastin Time (=aPTT) Prothrombin Time (Quick and International normalised ratio (INR)) |
| Enzymes | Aspartate Aminotransferase/ Glutamate-Oxaloacetate Transaminase (AST/GOT) Alanine transaminase(Glutamic Pyruvate Transaminase (ALT/GPT) Alkaline Phosphatase (AP/ALP) Creatine Kinase (CK) CK-MB if CK is elevated Lactic Dehydrogenase (LDH) |
| Substrates | Glucose Creatinine Blood urea nitrogen Bilirubin Total Bilirubin Direct Protein, Total C-Reactive Protein (CRP) Uric Acid Cholesterol, total High density lipoprotein (HDL) Cholesterol Calculated low density lipoprotein (LDL) Cholesterol Triglycerides |
| Electrolytes | Calcium<br>Sodium<br>Potassium |

Table 5.2.3: 2 Safety laboratory tests (cont'd)

| Category | Test name |
|---|---|
| Urinalysis (Stix) | Urine Nitrite |
| | Urine Protein |
| | Urine Glucose |
| | Urine Ketone |
| | Urobilinogen |
| | Urine Bilirubin |
| | Urine RBC/Erythrocyte |
| | Urine WBC/Leukocytes |
| | Urine pH |
| | Urine albumin (microalbumin urine test) (roll-over visit only) |
| Urine-Sediment | Urine Sediment Bacteria |
| (microscopic examination) | Urine Cast in Sediment |
| (if urine analysis abnormal) | Urine Squamous Epith Cells |
| , | Urine Sediment Crystals, Unspecified |
| | Urine Sediment red blood cell count (RBC)/Erythrocytes |
| | Urine Sediment white blood cell count (WBC)/Leucocytes |

# 5.2.4 Electrocardiogram

The 12-lead ECGs (I, II, III, aVR, aVL, aVF, V1-V6) will be recorded after the patients have rested for at least 5 minutes in a supine position. Electrode placement will be performed according to the method of Wilson, Goldberger and Einthoven. The ECGs will be evaluated by the study physician investigator or designee. ECGs may be repeated for quality reasons and the repeat tracing may be used for analysis. Additional ECGs may be collected by the investigator for safety reasons. Abnormal ECG recordings will be noted, and clinically relevant abnormal findings will be reported as AEs by the investigator. Any ECG abnormalities will be carefully monitored and if necessary medically treated.

ECG recordings will be obtained from roll-over visit and every 24 weeks, until study end including Extended EOT visit and Extended EOS visit

ECG measurements should, if possible, always precede blood sampling to avoid impact of sampling on the ECG results.

Signed and dated printouts of either ECG tracings or electronic ECG reports will be kept in the subject's/patient's medical file.

# 5.2.5 Assessment of other safety parameters

#### Vital signs

Vital signs include blood pressure (BP), pulse rate (PR), respiratory rate (RR), and oral or tympanic body temperature.

Systolic and diastolic BP as well as PR (by palpation, counted for 1 minute) will be measured after 5 minutes of rest in the supine position. (cf. Flow Chart for time points).

Measurements of vital signs should, if possible, always precede blood sampling to avoid impact of sampling on the results of vital signs.

## Medical examination

Complete physical examination will include vital sign assessment and general appearance as well as evaluation of all organ systems (eyes, ears, nose, mouth, and throat, neck, respiratory, cardiovascular, chest, gastrointestinal, lymphatic, musculoskeletal, skin, neurologic and psychiatric). Targeted physical examination will include vital sign assessment and evaluation of organ systems associated with AE(s) symptoms or laboratory abnormalities.

The medical examination carried out at the initial roll-over visit, will include documentation of patient information, informed consent, demographics including weight and waist circumference, smoking and alcohol history, relevant medical history and concomitant medication, review of inclusion/exclusion criteria, review of vital signs, 12-lead ECG and laboratory, and a complete physical examination.

## Local tolerability

Local tolerability at the administration site of the subcutaneous injection will be assessed by the investigator according to "swelling", "induration", "heat", "redness", "pain", or "other findings".

## 5.3 OTHER

## 5.3.1 Other endpoint(s)

Not applicable

## 5.3.2 Other assessment(s)

Not applicable

# 5.3.3 Pharmacogenomic evaluation

No pharmacogenetic samples will be collected in this study, as those samples will be available from the preceding trial.

# 5.4 APPROPRIATENESS OF MEASUREMENTS

The majority of measurements performed during this trial are standard measurements and will be performed in order to monitor safety aspects and to determine efficacy, PK and PD parameters in an appropriate way.

The scheduled measurements are appropriate to see drug induced changes in vital signs, standard laboratory values and ECG. These safety measurements standard and accepted for

#### Proprietary confidential information.

evaluation of safety and tolerability of an s.c. drug, and they are widely used in this kind of study.

The PK parameters and measurements outlined in Section 5.5 are generally used as measurements to assess drug exposure.

The efficacy endpoints are standard for assessment of patients with moderate to severe psoriasis. In addition, a number of exploratory PD measures (biomarkers) are also incorporated in this CTP. As these biomarkers have not been validated as prognostic measures, they may be analysed selectively and may not be included in the clinical trial report.

# 5.5 DRUG CONCENTRATION MEASUREMENTS AND PHARMACOKINETICS

Time points for dosing, PK and ADA sampling are listed in <u>Flow Chart.</u> Date and exact clock time of administration as well as pharmacokinetic and ADA sampling time points will be recorded. They will be documented in the CRFs by the medical personnel.

#### 5.5.1 Pharmacokinetic endpoint(s)

PK samples will serve to determine the following endpoints:

• steady state trough concentrations of BI 655066.

Individual concentration-time data with descriptive statistics for trough concentrations will be presented in the CTR. If deemed necessary, further appropriate pharmacokinetic parameters might be calculated.

Pharmacokinetic data may additionally be analysed using population pharmacokinetic approach. For this purpose data may also be combined with data from other trials. Modelling activities will be planned and documented separately.

#### 5.5.2 Methods of sample collection

#### 5.5.2.1 Plasma sampling for pharmacokinetic analysis

For the quantification of analyte plasma concentrations, approximately 2.5 mL of blood will be taken from a forearm vein into a K<sub>3</sub>EDTA (ethylendiaminetetraacetic acid) anticoagulant blood-drawing tube at the time points listed in Flow Chart under PK sampling.

Mix the K<sub>3</sub>EDTA-anticoagulated blood samples gently and place on ice until centrifugation at approximately +4°C. The blood should be centrifuged to produce plasma as soon as possible after collection, but not later than 30 minutes after withdrawal. Centrifugation will last for approximately 10 minutes (at 2000 x g to 4000 x g) at approximately +4°C. Two aliquots of EDTA plasma samples will be obtained in two polypropylene cryotubes. The two aliquots should contain approximately 0.5 mL of plasma each. Until shipment on dry ice to the analytical laboratory, the plasma samples will be stored at -20°C or below at the clinical

site and at the analytical laboratory until analysis. Both aliquots will be shipped (in separate shipments) to the assay laboratory for the determination of BI 655066. Both aliquots will be stored until the finalization of the clinical trial report and permission for sample disposal is provided. Samples will be shipped on dry ice sufficient for 3 days transit.

#### 5.5.2.2 Plasma sampling for assessment of anti-drug antibody

For the assessment of anti-drug antibody, approximately 2.5 mL of blood will be taken from a forearm vein into a K<sub>3</sub>EDTA anticoagulant blood-drawing tube at the time points listed in the Flow Chart under ADA.

Mix the K<sub>3</sub>EDTA-anticoagulated blood samples gently and place on ice until centrifugation at approximately +4°C. The blood should be centrifuged to produce plasma as soon as possible after collection, but not later than 30 minutes after withdrawal. Centrifugation will last for approximately 10 minutes (at 2000 x g to 4000 x g) at approximately +4°C. Two aliquots of EDTA plasma samples will be obtained in two polypropylene cryotubes. Both aliquots should contain approximately 0.5 mL of plasma each. Until shipment on dry ice to the analytical laboratory, the plasma samples will be stored at -20°C or below at the clinical site and at the analytical laboratory until analysis. Both aliquots will be shipped (in separate shipments) to the assay laboratory for the assessment of potential ADA to BI 655066. The ADA sample aliquots will be banked for possible/ additional ADA characterization in the future. Samples will be shipped on dry ice sufficient for 3 days transit.

#### 5.5.3 Analytical determinations

BI 655066 concentrations will be determined by a validated Enzyme Linked Immunosorbent Assay (ELISA).

The presence of ADA to BI 655066 will be assessed via a tiered approach using a validated electrochemiluminescence assay (screening, confirmatory, and titration analysis as appropriate). Samples that are confirmed positive will then be characterized in a validated neutralizing antibody (NAb) assay.

## 5.6 BIOMARKER(S)

Biomarkers associated with psoriatic disease and the IL-23 pathway will be assessed in plasma and serum from psoriasis patients, post treatment with BI 655066.

Blood samples (serum and plasma) will be collected at time points indicated in Flow Chart for the analysis of biomarkers. After completion of the study these samples may be used for not yet specified non-genetic biomarker analyses associated with autoimmune diseases as well as method development and evaluation. Samples will be stored for a maximum of 3 years (under consideration of local legislation) upon signature of the final study report.

#### 5.6.1 Endpoints based on biomarker(s)

Serum and plasma will be collected to assess changes in protein levels of disease specific markers such as but not limited to  $\beta$  defensin 2, neutrophil gelatinase associated lipocalin (NGAL), and S-100 proteins (A7, A8, A12) post treatment with BI 655066. These biomarkers are considered exploratory biomarkers and respective assays will need to be qualified to meet the required performance criteria.

## 5.6.2 Methods of sample collection

For the assessment of soluble protein biomarkers in serum, approximately 8 ml of blood will be collected from a forearm vein in a serum separation tube at time points indicated in the Flow Chart. The blood will be thoroughly mixed with clotting activation agent by inverting the tube not less than five times and will be allowed to clot for 30 minutes with the tube standing upright. The tube is then centrifuged at 1500 to 2000 x g for 15 minutes until clot and serum are separated by a well formed barrier. The serum will then be aliquoted in at least 6 aliquots (in polypropylene tubes) of at least 500 µl and should be frozen immediately at -20°C or below until shipment on dry ice to the analytical laboratory.

For the assessment of soluble protein biomarkers in plasma, approximately 8 ml of blood will be collected from a forearm vein in a potassium -EDTA (ethylendiaminetetraacetic acid)-anticoagulant blood drawing tube at the time points indicated in the Flow Chart. Tube content will be mixed immediately by gently inverting the tube at least 8 to 10 times and tube will then be transferred into an ice bath until centrifugation. The EDTA-anticoagulated blood sample will be centrifuged within 30 minutes after collection (intermittent storage in ice water or on ice). Centrifugation will last for about 10 minutes at 2000-4000 x g at 4-8°C until cells and plasma are well separated. After centrifugation, the EDTA plasma will be aliquoted in at least 6 aliquots (in polypropylene tubes) of at least 500  $\mu$ l and will be frozen immediately at -20°C or below.

# 5.6.3 Analytical determinations

Characteristics of the analytical methods for the analysis of serum and plasma biomarkers will be given in detail in the clinical trial report or in an accompanying technical/biomarker report.

#### 5.7 PHARMACODYNAMICS

Serum and plasma will be collected to assess changes in the levels of disease specific markers such as but not limited to  $\beta$  defensin 2, neutrophil gelatinase associated lipocalin (NGAL), and S-100 proteins (A7, A8, A12).

#### 5.7.1 Pharmacodynamic endpoints

Cf. section 5.6.1.

# 5.7.2 Methods of sample collection

Cf. section 5.6.2.

#### 5.8 PHARMACOKINETIC - PHARMACODYNAMIC RELATIONSHIP

No formal analysis of pharmacokinetic/pharmacodynamic relationships is planned.

If the data suggest a pharmacokinetic/pharmacodynamic relationship of special parameters, e.g. PASI, a detailed analysis may be performed.

Correlation between drug concentration and response may be made if adequate data are available. In addition, exploratory correlations may also be made between drug concentration and AEs.

Data may also be used to develop pharmacokinetic/pharmacodynamic models using nonlinear mixed effect modelling techniques, if feasible. For this purpose data may also be combined with data from other trials. Modelling activities will be planned and documented separately according to internal and external guidelines and SOP.


# 6. INVESTIGATIONAL PLAN

#### 6.1 VISIT SCHEDULE

All subjects have to adhere to the visit schedule as specified in <u>Flow Chart</u>. Any missed appointments should be re-scheduled as soon as possible. If any visit has to be rescheduled, subsequent visits should follow the original visit date scheduled. The investigator/sponsor could decide to arrange an unscheduled visit if deemed necessary (e.g. for safety follow-up reasons).

For detailed description of the trial procedures, please refer to Flow Chart.

In general, if several measurements including venipuncture are scheduled for the same point of time, venipuncture should, if possible, be the last of the measurements due to its mild discomfort to the patient and possible influence on physiologic parameters.

#### 6.2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS

# 6.2.1 Screening and run-in period(s)

Patients in the 1311.2 trial that fulfil the criteria for roll over, either by response < PASI<sub>50</sub> between week 24 and week 44, or completing the entire preceding trial reaching week 48 according to protocol, will be asked to participate in this open label extension trial. Upon their agreement, they will immediately enter the treatment phase. Therefore, no screening or run-in procedures are defined in this protocol.

#### 6.2.2 Treatment period(s)

#### 6.2.2.1 Rollover visit - Extended visit 1

After the approval of this protocol amendment in each respective country, all patients will follow Flow Chart (Extended dosing period) and receive 90mg BI 655066 subcutaneously at their Extended visit 1 (EV1). From EV1 onwards, BI655066 will be administered subcutaneously every 12 weeks during the trial. At EV2, if there is inadequate response, defined as <PASI<sub>90</sub>, the dose should be increased to 180mg for the remainder of the trial.

For ongoing patients from under the previous amendment (Pre-Extended Dosing Period, see Figure 3.1.3), EV1 should be conducted at the following time points:

- 1. For ongoing patients with ≥12 weeks since the EOT visit: Conduct EV1 as soon as possible
- 2. For ongoing patients still undergoing treatment or with <12 weeks since the EOT visit: Conduct EV1 at the time of the next scheduled treatment or follow up visit (note: EV1 should not be conducted at the time point of Visit 2 under the previous protocol, patients with Visit 2 as their next scheduled visit should have their EV1 replacing their Visit 3 instead)

Patients completing their EOS of 1311.2 and rolling over after approval of this protocol amendment, is immediately entering the Extended dosing period at EV1 of this trial. Eligible patients from 1311.2 who sign the informed consent for trial 1311.13, should preferably have Extended visit 1 of trial 1311.13 performed on the same day as the last visit in 1311.2, or within an interim period of up to 6 weeks thereafter.

Assessments performed at EOS in the previous trial do not have to be repeated at Extended visit 1 in this trial, if performed as combined visits. If EV1 is performed as a separate visit to 1311.2 EOS, all EV1assessments should be performed, but specific assessments are only required at EV1 for patients that are having EV1 as their first 1311.13 visit, see Flow Chart for further instructions.

Written informed consent in accordance with GCP and local legislation must be obtained prior to any study related procedure taking place. If not performed as combined visits, informed consent must therefore be signed before the roll-over visit due to lab sampling fasting at EV1 in trial 1311.13.

Review of the following inclusion/exclusion criteria will be based on the last available lab result from previous trial, at the time of roll-over, and needs to be re-assessed as soon as 1311.2 EOS/1311.13 roll-over visit results are available:

• Inclusion criteria 3 (Negative serum β-Human Chorionic Gonadotropin (β-HCG)) Exclusion criteria 8 (Any clinically significant laboratory abnormalities)

Check consistency in medical history with the data obtained at visit 1 of the previous trial. All changes in medical history must be documented as adverse events and will be followed up as such during this trial.

Re-record ongoing adverse events/concomitant medications from the previous trial and record any adverse events/concomitant medications that may have started between the two trials, in the event that the 6 week time-window between trials was used.

All patients will be administered 90 mg BI 655066 s.c. at Extended visit 1.

#### 6.2.2.2 Extended Dosing Period

After 12 weeks, if there is a lack of response, defined as response below PASI<sub>90</sub> at Extended visit 2, the dose should be increased to 180 mg, and 180 mg dosing will occur every 12 weeks until Extended EOT.

Self-administered patient questionnaire (DLQI) should be completed by the patient before any other visit assessments or treatments.

For detailed description of the trial procedures, please refer to Flow Chart.

#### 6.2.3 End of trial and Extended follow-up period

Trial 1311.13 is an open label extension trial which was set up in order to assess the long term safety and efficacy of Risankizumab (BI 655066) in patients with plaques psoriasis who have completed the phase 2 trial 1311.2. Moreover, this trial was meant to offer patients continuous treatment with Risankizumab until the marketing approval and availability of Risankizumab in the respective participating countries.

In the course of the acquisition of Risankizumab by Abbvie and the transition of responsibilities from BI to Abbvie it is planned to transfer the patients who are treated in 1311.13 into M15-997 which is sponsored and conducted by Abbvie. M15-997 is an open label extension trial in which patients who have completed one of the Risankizumab pivotal trials in the indication of plaques psoriasis receive 150 mg Risankizumab every 12 weeks.

For patients who discontinue study medication before Extended end of treatment (for any reason), or before approval of this amendment and start to rollover patients to the M15-997 from 01-May-2018 an early Extended EOT visit should be scheduled. If the decision to discontinue study participation is taken at a regular study visit, the visit should be turned into an Extended EOT visit. If the decision to discontinue study participation is taken in between study visits, an Extended EOT visit is to be scheduled at the earliest convenience and by the latest at the next upcoming visit according to the Flow Chart. This early Extended EOT visit will include the same procedures as the normal EOT, and the patient will subsequently enter a follow up period of 12 weeks, until a final Extended EOS visit is performed. If the decision to discontinue is taken in the Extended follow up period, the Extended EOS visit is to be scheduled at the earliest convenience. The procedures described at Extended EOS will be performed and the information will be recorded in the CRFs.

The end of study procedures are listed in Flow Chart.

#### 6.2.3.1 Vital status

In case of early discontinuation, information should be collected to differentiate between patients lost to follow-up (investigator not able to contact the patient despite multiple attempts) versus patients the investigator was able to contact who elected to discontinue study participation for any reason. Patients will be asked to give consent to be contacted (or for their primary care physician to be contacted) by the study team to obtain vital status information preferably at the time of study entry. This consent must be documented in the patient notes. Patient's vital status, including cause of death, will be collected every 12 months from Extended EOS until the last patient completes the regular scheduled Extended EOS. Vital status data will be collected in the eCRFs.

All clinically significant abnormal values (including laboratory parameters) will be followed up using the appropriate tests until a return to a medically acceptable level is achieved. AEs persisting after trial completion must be followed up, until they have normalised or been sufficiently characterised.

# 7. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

#### 7.1 STATISTICAL DESIGN - MODEL

This is a double arm extension trial of patients treated with BI 655066 after participation in a clinical trial of BI 655066. Descriptive statistical models include a responder analysis (e.g., achieving PASI<sub>90</sub>, sPGA of clear or almost clear, etc.), time to loss of response (e.g., achieving PASI<sub>90</sub>, sPGA of clear or almost clear, etc.), time to AESI, and time to antibody development formation. No statistical testing will be done.

#### 7.2 NULL AND ALTERNATIVE HYPOTHESES

The primary hypothesis is that BI 655066 will sustain effectiveness without emergent safety issues during the extended visit period. This will be characterized descriptively. There is no formal statistical hypothesis testing in this study.

#### 7.3 PLANNED ANALYSES

The descriptive analyses will be based on proportions of patients achieving a response (e.g., achieving PASI<sub>90</sub>, sPGA of clear or almost clear, etc.), Kaplan Meier empirical survival curves to describe patterns of event incidence, and cumulative event rates at critical timepoint.

The study is designed to gain as much exposure as possible with adequate documentation of safety, efficacy, and antibody emergence.

For all analyses, baseline refers to the baseline value in the 1311.2 study.

# 7.3.1 Primary analyses

The achievement of PASI90 at week 48 in the Extended dosing period is the primary efficacy endpoint, which is a binary variable.

For primary safety, the overall incidence rates of AEs, drug related AEs, and SAEs will be calculated.

#### 7.3.2 Secondary analyses

The same methods as discussed for the primary analyses will be used to analyse all binary secondary and other endpoints, which include achievement of PASI50 / PASI75 / PASI90 / PASI100 at all Extended dosing period visits where PASI is collected and achievement of sPGA of clear or almost clear at all Extended dosing period visits where sPGA is collected.

Time to loss of PASI<sub>50</sub> / PASI<sub>75</sub> / PASI<sub>90</sub> / PASI<sub>100</sub>, and time to loss of sPGA of clear or almost clear will be analysed using a Kaplan-Meier estimate.

Percent change from baseline in Pain-VAS for patients with non-zero baseline will be summarized descriptively at time points collected.

DLQI will be summarized descriptively at time points collected.

Additional information on these analyses will be provided in the trial statistical analysis plan.

# 7.3.3 Safety analyses

All subjects who received one dose of study drug will be included in the safety evaluation.

Safety analyses will focus on adverse events related to early discontinuation, immune suppression and injection site effects. AEs will be coded using the Medical Dictionary for Drug Regulatory Affairs (MedDRA). All AEs occurring up to 12 weeks after the last trial medication administration will be assigned to the treatment period for evaluation. The evaluation of adverse events will comprise various frequency tabulations. The additional analyses of pre-defined AESI will consider the frequency, intensity, time to first onset of the AE, duration of the AE and clinical consequences (e.g. study discontinuation).

Analysis of laboratory measures will similarly focus on hematologic measures of immune suppression. Descriptive statistics of laboratory values over time and for the difference from baseline will be provided. Frequency tables of changes with respect to the reference range between baseline and last/worst value on treatment and patients with possible clinically significant abnormalities will also be presented.

Immunogenicity will be evaluated in terms of time to antibody emergence starting from the time of first exposure to BI 655066 in either 1311.2 or 1311.13. This will be analysed using a Kaplan-Meier estimate.

Safety will also be assessed by evaluation of vital signs (BP, PR, RR, oral or tympanic body temperature) and local tolerability.

#### 7.3.4 Interim analyses

Results will be analysed periodically by the sponsor and DMC in order to review the accumulating safety data of BI 655066 in psoriasis.

# 7.3.5 Pharmacokinetic analyses

Individual concentration-time data with descriptive statistics for trough concentrations will be presented in the clinical trial report.

Population pharmacokinetic/pharmacodynamic analysis, if performed, will be reported separately.

#### 7.3.6 Pharmacodynamic analyses

Serum/plasma biomarkers will be summarized over time and correlated with clinical endpoints (i.e. PASI, PGA).

# 7.3.7 Pharmacogenomic analyses

Not applicable.

#### 7.4 HANDLING OF MISSING DATA

Use of inappropriate concomitant medication to treat psoriasis will be considered as failure when deriving response variables, e.g. PASI<sub>90</sub>.

Further details on the handling of missing data will be provided in the Trial Statistical Analysis Plan.

#### 7.5 RANDOMISATION

There is no randomisation for this study. All patients will be assigned to the same regimen and dose of BI 655066, regardless of the treatment and dose received in the 1311.2 study.

# 7.6 DETERMINATION OF SAMPLE SIZE

The sample size is determined by the completion of previous trial and the consenting for the extension.


# 8. INFORMED CONSENT, DATA PROTECTION, TRIAL RECORDS

The trial will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, in accordance with the International conference on harmonisation (ICH) Harmonised Tripartite Guideline for Good Clinical Practice (GCP) and relevant BI Standard Operating Procedures (SOPs). Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician of the patient.

The investigator should inform the sponsor immediately of any urgent safety measures taken to protect the study subjects against any immediate hazard, and also of any serious breaches of the protocol/ICH GCP.

The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract. As a general rule, no trial results should be published prior to finalisation of the Clinical Trial Report.

<u>Insurance Cover:</u> The terms and conditions of the insurance cover are made available to the investigator and the patients via documentation in the ISF (Investigator Site File).

# 8.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This trial will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB) / Independent Ethics Committee (IEC) and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

Prior to patient participation in the trial, written informed consent must be obtained from each patient (or the patient's legally accepted representative) according to ICH GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional patient-information form retained by the investigator as part of the trial records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative.

The patient must be informed that his/her personal trial-related data will be used by Boehringer Ingelheim in accordance with the local data protection law. The level of disclosure must also be explained to the patient.

The patient must be informed that his / her medical records may be examined by authorised monitors (CML/CRA) or Clinical Quality Assurance auditors appointed by Boehringer Ingelheim, by appropriate IRB / IEC members, and by inspectors from regulatory authorities.

# 8.2 DATA QUALITY ASSURANCE

A quality assurance audit/inspection of this trial may be conducted by the sponsor or sponsor's designees or by IRBs/IECs or by regulatory authorities. The quality assurance

auditor will have access to all medical records, the investigator's trial-related files and correspondence, and the informed consent documentation of this clinical trial.

#### 8.3 RECORDS

Case Report Forms (CRFs) for individual patients will be provided by the sponsor, either on paper or via remote data capture. For drug accountability, refer to Section 4.1.8.

#### 8.3.1 Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

Data entered in the eCRFs that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the trial; also current medical records must be available.

For eCRFs all data must be derived from source documents.

#### 8.3.2 Direct access to source data and documents

The investigator / institution will permit trial-related monitoring, audits, IRB / IEC review and regulatory inspection, providing direct access to all related source data / documents. CRFs/eCRFs and all source documents, including progress notes and copies of laboratory and medical test results must be available at all times for review by the sponsor's clinical trial monitor, auditor and inspection by health authorities (e.g. Food and Drug Administration (FDA)). The Clinical Research Associate (CRA) / on site monitor and auditor may review all CRFs/eCRFs, and written informed consents. The accuracy of the data will be verified by reviewing the documents described in Section 8.3.1.

#### 8.4 LISTEDNESS AND EXPEDITED REPORTING OF ADVERSE EVENTS

#### 8.4.1 Listedness

To fulfil the regulatory requirements for expedited safety reporting, the sponsor evaluates whether a particular adverse event is "listed", i.e. is a known side effect of the drug or not. Therefore a unique reference document for the evaluation of listedness needs to be provided. For the BI 655066 this is the current version of the Investigator's Brochure (<u>U12-3042</u>). The current version of this reference document is to be provided in the ISF. No AEs are classified as listed for matching placebo, study design, or invasive procedures.

# 8.4.2 Expedited reporting to health authorities and IECs/IRBs

Expedited reporting of serious adverse events, e.g. suspected unexpected serious adverse reactions (SUSARs) to health authorities and IECs/IRBs, will be done according to local regulatory requirements. Further details regarding this reporting procedure are provided in the Investigator Site File.

#### 8.5 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this trial is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

Treatment data may be given to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated as a result of the trial need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB / IEC and the regulatory authorities i.e. the CA.

#### 8.6 COMPLETION OF TRIAL

The EC/competent authority in each participating EU member state needs to be notified about the end of the trial (last patient out, unless specified differently in <u>Section 6.2.3</u> of the CTP) or early termination of the trial.

# 9. REFERENCES

#### 9.1 PUBLISHED REFERENCES

- P06-11555 Filipe-Santos O, Bustamante J, Chapgier A, Vogt G, Beaucoudrey L de, Feinberg J, Jouanguy E, Boisson-Dupuis S, Fieschi C, Picard C, Casanova JL. Inborn errors of IL-12/23- and IFN-gamma-mediated immunity: molecular, cellular, and clinical features. Semin Immunol 2006. 18(6):347-361.
- R03-1207 A new scoring system to determine if clinically significant improvement has occurred in clinical trials that assess the effect of therapy on psoriasis (version 6, Aug 22, 2001). Medical Advisory Board of the National Psoriasis Foundation 2001
- R03-1208 NPF psoriasis score. Psoriasis Forum 2002. 8(2)
- R05-2548 Finlay AY, Khan GK. Dermatology Life Quality Index (DLQI) a simple practical measure for routine clinical use. Joint Ann Mtg of the British Association of Dermatologists and the Canadian Dermatology Association, Oxford, 6 10 Jul 1993 Clin Exp Dermatol 1994. 19:210-216.
- R08-1089 Lowes MA, Bowcock AM, Krueger JG. Pathogenesis and therapy of psoriasis. Nature 2007; 445(7130):866-873.
- R11-1204 Ghilardi N, Kljavin N, Chen Q, Lucas S, Gurney AL, Sauvage FJ de.
  Compromised humoral and delayed-type hypersensitivity responses in IL-23deficient mice. J Immunol 2004. 172:2827-2833.
- R11-1236 Meeran SM, Mantena SK, Meleth S, Elmets CA, Katiyar SK. Interleukin-12-deficient mice are at greater risk of UV radiation-induced skin tumors and malignant transformation of papillomas to carcinomas. Mol Cancer Ther 2006. 5(4):825-832.
- R11-1257 Nestle FO, Kaplan DH, Barker J. Mechanisms of disease: psoriasis. N Engl J Med 2009; 361(5):496-509.
- R11-1259 Menter A, Griffiths CEM. Psoriasis 2: current and future management of psoriasis. Lancet 2007; 370:272-284.
- R11-1261 Leon A, Nguyen A, Letsinger J, Koo J. An attempt to formulate an evidence-based strategy in the management of moderate-to-severe psoriasis: a review of the efficacy and safety of biologics and prebiologic options. Expert Opin Pharmacother 2007; 8(5):617-632.
- R11-1529 Gordon KB, Langley RG, Gottlieb AB, Papp KA, Krueger GG, Strober BE, et al. A phase III, randomized, controlled trial of the fully human IL-12/23/mAb briakinumab in moderate-to-severe psoriasis. J Invest Dermatol e-pub ahead of print 20 October 2011.

R11-4193 Ryan C, Leonardi CL, Krueger JG, Kimball AB, Strober BE, Gordon KB, et al. Association between biologic therapies for chronic plaque psoriasis and cardiovascular events: a meta-analysis of randomized controlled trials. JAMA 2011; 306(8):864-871. R12-1008 Iwakura Y, Nakae A, Saijo S, Ishigame H. The roles of IL-17A in inflammatory immune responses and host defense against pathogens. Immunol Rev 2008. 226:57-79. R12-1010 Reich K, Langley RG, Papp KA, Ortonne JP, Unnebrink K, Kaul M, Valdes JM. A 52-week trial comparing briakinumab with methotrexate in patients with psoriasis. N Engl J Med 2011. 365(17):1586-1596. Chackerian AA, Chen SJ, Brodie SJ, Mattson JD, McClanahan TK, Kastelein R12-1011 RA, Bowman EP. Neutralization or absence of the interleukin-23 pathway does not compromise immunity to mycobacterial infection. Infect Immun 2006. 74(11):6092-6099. Woodworth T et al.. Standardizing Assessment and Reporting of Adverse R13-3515 Effects in Rheumatology Clinical Trials II: the Rheumatology Common Toxicity Criteria v. 2.0. J Rheumatol 2007; 34:1401-14. R13-3518 Papp-KA, Griffiths-CEM, Gordon-K, Lebwohl-M, Szapary-PO, Wasfi-Y, Chan-D, Hsu-MC, Ho-V, Gishlain-PD, Strober-B, Reich-K. Long-term safety of ustekinumab in patients with moderate-to-severe psoriasis: final results from 5 years of follow-up. Br J Dermatol 2013; 168:844-854. R96-3541 Fredriksson T, Pettersson U. Severe psoriasis - oral therapy with a new retinoid. Dermatologica 1978; 157:238-244. Husni ME, Meyer KH, Cohen DS, Mody E, Oureshi AA R13-3802 The PASE questionnaire: pilot-testing a psoriatic arthritis screening and evaluation tool. J Am Acad Dermatol 57 (4), 581 - 587 (2007)

#### 9.2 UNPUBLISHED REFERENCES

- U12-3042 Investigator's Brochure BI 655066, Psoriasis, Crohn's Disease, Ankylosing Spondylitis, 1311.P1/1311.P2/1311.P3
- M14-0004 Manuscript: Anti-IL-23 monoclonal antibody BI 655066 in treatment of psoriasis: Safety, efficacy pharmacokinetics and biomarker results of a single rising dose, randomized, double-blind, placebo-controlled trial Submitted for publication


# 10. APPENDICES

#### 10.1 PASI SCORE DEFINITION AND INSTRUCTIONS

The PASI score is an established measure of clinical efficacy for psoriasis medications. (R96-3541)

To calculate the PASI score, the four main body areas are assessed: **head (h), trunk (t), upper extremities (u) and lower extremities (l).** These correspond to 10, 30, 20 and 40% of the total body area respectively.

The area of psoriatic involvement of these four areas (Ah, At, Au, and Al) is given a numerical value: 0 = no involvement, 1 = <10%, 2 = 10 to <30%, 3 = 30 to <50%, 4 = 50 to <70%, 5 = 70 to <90%, and 6 = 90 to 100% involvement.

The signs of severity, erythema (E), infiltration (I) and desquamation (D) of lesions are assessed using a numeric scale 0-4 where 0 is a complete lack of cutaneous involvement and 4 is the severest possible involvement; scores are made independently for each of the areas, h, t, u and l and represents a composite score for each area. An illustration of judging erythema follows: 0 = no erythema, 1 = slight erythema, 2 = moderate erythema, 3 = striking erythema, and 4 = exceptionally striking erythema.

The PASI score is calculated according to the following formula:

PASI = 0.1(Eh + Ih + Dh)Ah + 0.3(Et + It + Dt)At + 0.2(Eu + Iu + Du)Au + 0.4(El + Il + Dl)Al

# 10.2 STATIC PHYSICIAN'S GLOBAL ASSESSMENT (SPGA) OF THE NPF PSORIASIS SCORE (NPFPS)

The NPF Psoriasis Score (NPFPS) was devised by the National Psoriasis Foundation Medical

Advisory Board to address deficiencies inherit in the PASI, and to provide a dynamic, reproducible, and easy 5-component method to measure clinically significant improvement in trials of new or existing psoriatic therapies (<u>R03-1207</u>, <u>R03-1208</u>). The static Physician Global Assessment (sPGA) is one of five components of the NPFPS, and may be used independently (R03-1207, R03-1208).

The primary sPGA variable to be analysed will be the proportion of patients that are "clear or almost clear". This has been shown to correlate well with PASI75 or higher score.

For patients to be considered "clear," the average of the 3 components must be zero (with standard rounding rules, i.e., 0.333 rounds to 0) and the score for thickness must equal zero.

For patients to be considered "almost clear," the average of the 3 components must be 1 (with standard rounding rules, i.e., 1.333 rounds to 1) and each of the individual components must be less than 3 (in other words, each of the 3 components must be equal 0, 1, or 2).

Additionally, patients with an average of the 2 components equal to zero but with a thickness score of 1 will be considered as "almost clear."

# **Static Physician Global Assessment (averaged over all lesions)**

| 0 | clear | = cleared, except for residual discoloration |
|---|---|---|
| 1 | almost clear | = majority of lesions have individual scores for thickness (a), erythema (b) and scaling (c) that averages 1. |
| 2 | mild | = majority of lesions have individual scores for thickness (a), erythema (b) and scaling (c) that averages 2. |
| 3 | moderate | = majority of lesions have individual scores for thickness (a), erythema (b) and scaling (c) that averages 3. |
| 4 | marked | = majority of lesions have individual scores for thickness (a), erythema (b) and scaling (c) that averages 4. |
| 5 | severe | = majority of lesions have individual scores for thickness (a), erythema (b) and scaling (c) that averages 5. |

## (a) Thickness (averaged over all lesions)

0 = no evidence of plaque elevation

1 = minimal plaque elevation,  $\approx 0.25$  mm

 $2 = \text{mild plaque elevation}, \approx 0.5 \text{ mm}$ 

- $3 = \text{moderate plaque elevation}, \approx 0.75 \text{ mm}$
- $4 = \text{marked plaque elevation}, \approx 1 \text{ mm}$
- 5 = severe plaque elevation,  $\approx 1.25$  mm or more

Thickness in the sPGA may be graded with the aid of a reference card, which has embossed elevations ranging from 0 to 1.25 mm that increase linearly at 0.25 mm increments corresponding to varying levels of thickness (0-5) for each target lesion. The dermatologist should select 3 or more representative lesions (e.g., lesions not on the face, scalp, intertriginous areas or only on elbows or knees) at the time of the visit and measure their thickness. These can be averaged to derive the thickness score. The investigator should assess the average degree of thickness and then select the number that most represents this. For any assessments that fall half way between any two numbers on the scale, the investigator will be told to always round up to the higher number. This would result in then the following implied range: 0 = 0 to < 0.125 mm,  $1 = \ge 0.125$  to < 0.375 mm,  $2 = \ge 0.375$  to < 0.625mm,  $3 = \ge 0.625$  to < 0.875mm,  $4 = \ge 0.875$  to < 1.25mm and  $5 = \ge 1.25$ mm.

#### (b) Erythema (averaged over all lesions)

0 = no evidence of erythema, hypo- or hyper-pigmentation may be present

- 1 = faint erythema
- 2 = light red coloration
- 3 = moderate red coloration
- 4 = bright red coloration
- 5 =dusky to deep red coloration

#### (c) Scaling (averaged over all lesions)

- 0 = no evidence of scaling
- 1 = minimal; occasional fine scaling over less than 5% of the lesion
- 2 = mild; fine scaling predominates
- 3 = moderate; coarse scaling predominates
- 4 = marked; thick, non-tenacious scaling predominates
- 5 = severe; very thick tenacious scaling predominates

# 10.3 PAIN VISUAL ANALOG SCALE (VAS)

If a patient has psoriatic arthritis, the patient will assess their psoriatic arthritis at each protocol defined time point. A global estimate of pain caused by joint disease will be estimated by the patient's response to the question: "The very left end of the scale is equivalent to "no pain" at all whereas the right end of the scale is equivalent to "worst possible pain". How much pain have you had because of your illness in the past week?" Response is captured using a VAS (range 0 to 100, where 100 is highest severity) and results will be summarized.

#### 10.4 DERMATOLOGY LIFE QUALITY INDEX

DLQI is a subject-administered,10-question, validated, quality of life questionnaire that covers 6 domains including symptoms and feelings, daily activities, leisure, work and school, personal relationships and treatment. Response categories include "not relevant" (score of 0), "not at all" (score of 0), "a little" (score of 1), "a lot" (score of 2) and "very much" (score of 3). Question 7 is a "yes"/ "no" question where "yes" is scored as 3.

The DLQI will be analysed under six headings as follows (R05-2548):

| Domain | Question Number | Score |
|------------------------|-------------------|-----------------|
| Symptoms and feelings | Questions 1 and 2 | Score maximum 6 |
| Daily activities | Questions 3 and 4 | Score maximum 6 |
| Leisure | Questions 5 and 6 | Score maximum 6 |
| Work and school | Question 7 | Score maximum 3 |
| Personal relationships | Questions 8 and 9 | Score maximum 6 |
| Treatment | Question 10 | Score maximum 3 |

DLQI total score is calculated by summing the scores of each question resulting in a range of 0 to 30 where 0-1 = no effect on subject's life, 2-5 = small effect, 6-10 = moderate effect, 11-20 = very large effect, and 21-30 = extremely large effect on subject's life. The higher the score, the more the quality of life is impaired. If the answer to one question in a domain is missing, that domain is treated as missing. If 2 or more questions are left unanswered (missing), DLQI total score is treated as missing. A 5-point change from baseline is considered a clinically important difference.

# 10.5 PSORIATIC ARTHRITIS SCREENING AND EVALUATION TOOL

If a patient has psoriatic arthritis or if psoriatic arthritis is suspected at the roll-over visit, the psoriatic arthritis screening and evaluation (PASE) questionnaire should be performed. It will then be measured once per year until study end. The PASE questionnaire is a self-administered tool that can be used to screen for psoriatic arthritis among patients with psoriasis. PASE can distinguish between symptoms of psoriatic arthritis and osteoarthritis (R13-3802).

Psoriatic Arthritis Screening and Evaluation (PASE) Questionnaire

Please circle or mark ONLY ONE of the five choices on the following 15 questions. The answers to these questions will help us better understand your symptoms. This should take about 5 to 6 minutes to complete. Thank you for your time.


| Symptoms subscale | Strongly<br>disagree | Disagree | Neutral | Agree | Strongly agree |
|---|---|---|---|---|---|
| 1. I feel tired for the most of the day | 1 | 2 | 3 | 4 | 5 |
| 2. My joints hurt | 1 | 2 | 3 | 4 | 5 |
| 3. My back hurts | 1 | 2 | 3 | 4 | 5 |
| 4. My joints become swollen | 1 | 2 | 3 | 4 | 5 |
| 5. My joints feel "hot" | 1 | 2 | 3 | 4 | 5 |
| 6. Occasionally, an entire finger or toe becomes swollen, making it look like a "sausage" | 1 | 2 | 3 | 4 | 5 |
| 7. I have noticed that the pain in my joints moves from one joint to another, e.g. my wrist will hurt for a few days then my knee will hurt and so on | 1 | 2 | 3 | 4 | 5 |
| Symptom Score (Max 35) | Add scores | for questions | s 1-7 and writ | e next to A | A. |
| Function subscale | Strongly disagree | Disagree | Neutral | Agree | Strongly agree |
| 8. I feel that my joint problems have affected my ability to work | 1 | 2 | 3 | 4 | 5 |
| 9. My joint problems have affected my ability to care for myself, e.g. getting dressed or brushing my teeth | 1 | 2 | 3 | 4 | 5 |
| 10. I have had trouble wearing rings on my fingers or my watch | 1 | 2 | 3 | 4 | 5 |
| 11. I have had trouble getting into or out of a car | 1 | 2 | 3 | 4 | 5 |
| 12. I am unable to be as active as I used to be | 1 | 2 | 3 | 4 | 5 |
| 13. I feel stiff for more than two hours after waking up in the morning | 1 | 2 | 3 | 4 | 5 |
| 14. The morning is the worst time of the day for me | 1 | 2 | 3 | 4 | 5 |
| 15. It takes me a few minutes to get moving to the best of my ability, any time of the day | 1 | 2 | 3 | 4 | 5 |
| Function Score (Max 40) | Add scores | for questions | s 8-15 and wr | ite next to B | В. |
| Total PASE Score (Max 75) | Add scores | in boxes A a | nd B and wri | te next to C | C. |

#### 10.6 CLINICAL EVALUATION OF LIVER INJURY

#### 10.6.1 Introduction

Alterations of liver laboratory parameters, as described in <u>Section 5.2.2.1</u> (Adverse Events of Special Interest), are to be further evaluated using the following procedures:

#### 10.6.2 Procedures

Repeat the following laboratory tests: ALT, AST, and bilirubin (total and direct) - within 48 to 72 hours and provide additional blood sample to the central laboratory for automatic reflex testing of the below listed laboratory parameters. Only in case whereby the central laboratory is not immediately available (e.g. if the logistics are such that the patient's repeat specimen would not reach the central laboratory in a reasonable timeframe), ALT, AST, and bilirubin (total and direct) will be evaluated by local laboratory and results are made available to the investigator and to BI as soon as possible. If in such a case ALT and/or AST >3 fold ULN combined with an elevation of total bilirubin >2 fold ULN are confirmed, results of the laboratory parameters described below must be made available to the investigator and to BI as soon as possible.

#### In addition,

- o obtain a detailed history of current symptoms and concurrent diagnoses and medical history according to the "DILI checklist" provided in the ISF
- obtain history of concomitant drug use (including non-prescription medications, herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets according to the "DILI checklist" provided in the ISF;
- obtain a history of exposure to environmental chemical agents (consider home and work place exposure) according to the "DILI checklist" provided in the ISF;

and report these via the CRF.

#### Clinical chemistry

alkaline phosphatase, albumin, PT or INR, CK, CK-MB, ceruloplasmin,  $\alpha$ -1 antitrypsin, transferrin, amylase, lipase, fasting glucose, cholesterol, triglycerides

# Serology

Hepatitis A (Anti-IgM, Anti-IgG), Hepatitis B (HbsAg, Anti-HBs, DNA), Hepatitis C (Anti-HCV, RNA if Anti-HCV positive), Hepatitis D (Anti-IgM, Anti-IgG), Hepatitis E (Anti-HEV, Anti-HEV IgM, RNA if Anti-HEV IgM positive), Anti-Smooth Muscle antibody (titer), Anti-nuclear antibody (titer), Anti-LKM (liver-kidney microsomes) antibody, Anti-mitochondrial antibody

Hormones, tumormarker TSH

Haematology
Thrombocytes, eosinophils

- o Provide abdominal ultrasound to rule out biliary tract, pancreatic or intrahepatic pathology, e.g. bile duct stones or neoplasm.
- o Initiate close observation of subjects by repeat testing of ALT, AST, and total bilirubin (with fractionation by total and direct) at least weekly until the laboratory ALT and / or AST abnormalities stabilize or return to normal, then according to the protocol. Depending on further laboratory changes, additional parameters identified e.g. by reflex testing will be followed up based on medical judgement and Good Clinical Practices (GCP).

30 January 2018

Boehringer Ingelheim BI Trial No.: 1311.13

Doc. No.: c02318676-08

Trial Protocol


# SEVERITY OF AE AS DESCRIBED IN THE RHEUMATOLOGY COMMON TOXICITY CRITERIA V. 2.0 10.7

| Asympto transient Short du | | z - Iviouciaic | 3 - Severe | 4 - Includes Lile |
|---|---|---|---|---|
| Asyı<br>trans | | | | Threatening |
| Lans | Asymptomatic, or | Symptomatic | Prolonged symptoms, | At risk of death |
| | Islent | Direction (1 ) works | reversible, major | Carbotontiol discolative |
| | Short duration (< 1 | Duration (1–2 weeks) | runctional impairment | Substantial disability, |
| week) | ck) | Alter lifestyle | Prescription meds/partial | especially if permanent. |
| 9 oN | No change in life style | occasionally | relief | Multiple meds |
| Nor | No medication or over | Meds relieve. (may be | May be hospitalized < | Hospitalization > 24h |
| the c | the counter medication | prescription), | 24h | Study drug discontinued |
| (OTC) | () | Study drug continued | Temporary study drug | |
| | | | discontinuation, or/and | |
| | | | dose reduced | |
| A. ALLERGIC/IMMUNOLOGIC | OGIC | | | |
| A1. Allergic Tran | Transient rash; drug | Generalised urticaria | Symptomatic | Anaphylaxis, laryngeal/ |
| reaction/hyper- | fever < 38°C: transient | responsive to meds; or | bronchospasm, requiring | pharyngeal oedema, |
| sensitivity (including asyn | asymptomatic | drug fever $> 38^{\circ}$ C, or | meds; symptomatic | requiring resuscitation |
| drug fever) bron | bronchospasm | reversible bronchospasm | urticaria persisting with | |
| | | | meds, allergy related | |
| | | | oedema/angioedema | |

© 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. Proprietary confidential information.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

Trial Protocol


| A. ALLERGIC/IMMUNOLOGIC A2. Autoimmune Serologic or other evidence of autoimmune reaction, but patient asymptomatic: all organ function normal and no treatment is required | an | | Canses major organ |
|---|---|---|---|
| oimmune | an | | Canses major organ |
| | an | function of a major organ | Causes major organ |
| autoimmune reaction, but patient asymptomatic: all orgination normal and intreatment is required | an | function of a major organ | dysfunction, |
| but patient asymptomatic: all org function normal and 1 treatment is required | | or tovicity requiring short | or progressive, not |
| asymptomatic: all org<br>function normal and 1<br>treatment is required | | or coalcuty requiring smort | reversible, or requires |
| function normal and 1 treatment is required | | term immunosuppressive | long term administration |
| treatment is required | d no ımmunosuppressive | treatment (e.g. transient | of high dose |
| (P a vitilian) | ed drugs (e.g. | colitis or anaemia) | immunosuppressive |
| (c.g. v muse) | hypothyroidism) | | therapy |
| A3. Rhinitis (includes Transient, non- | Prescription med. | Corticosteroids or other | NA |
| sneezing, nasal prescription meds | required, | prescription med. with | |
| stuffiness, post-nasal relieve | slow | persistent disabling | |
| discharge) | | symptoms such as | |
| | | impaired exercise | |
| | | tolerance | |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

o.: c02318676-08

Trial Protocol


| 3 - Severe 4 - Includes Life Threatening | | Prolonged; symptoms Major organ dysfunction, only partially relieved by requires long-term high- | meds; parenteral dose immunosuppressive corticosteroids required therapy | Generalised, parenteral Prolonged, | or/and short duration | hospitalisation | | | maintenance prescription required; parenteral meds |
|---|---|---|---|---|---|---|---|---|---|
| 2 - Moderate | | Symptomatic, slow response to meds (e.g. | oral corticosteroids) | Symptomatic, slow | oral corticosteroids) | | | Transient, but | symptomatic or recurrent, responds to meds |
| 1 - Mild | LOGIC | Transient, non-<br>prescription meds | relieve | Localised, not requiring | response to meds; | cutaneous | | Transient, | asymptomatic |
| | ALLERGIC/IMMUNOLOGIC | A4. Serum sickness | | A5. Vasculitis | | | B. CARDIAC | B1. Arrhythmia | |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| B. CARDIAC | | | | |
| B2. Cardiac function | Asymptomatic decline | Asymptomatic decline of Congestive heart failure | Congestive heart failure | Severe or refractory CHF |
| decreased | in resting ejection | resting ejection fraction $\geq$ (CHF) responsive to | (CHF) responsive to | |
| | fraction by $> 10\%$ , but | 20% of baseline value | treatment | |
| | < 20% of baseline value | | | |
| B3. Edema | Asymptomatic (e.g. 1+ | Symptomatic (e.g. 2+ | Symptoms limiting | Anasarca; no response to |
| | feet/calves), self- | feet/calves), requires | function (e.g. 3+ | treatment |
| | limited, no therapy | therapy | feet/calves, $2+$ thighs), | |
| | required | | partial relief with | |
| | | | treatment, prolonged | |
| B4. Hypertension | Asymptomatic, | Recurrent or persistent | Symptomatic increase > | Hypertensive crisis |
| (new onset or | transient increase by > | increase $> 150/100$ or by | 150/100 > 20 mm Hg, | |
| worsening) | 20 mm Hg (diastolic), | > 10 mmHg (diastolic), | persistent, requiring | |
| | or to $> 150/100$ if | requiring and responding | multi-agent therapy, | |
| | previously normal, no | readily to treatment | difficult to control | |
| | therapy required | | | |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| B. CARDIAC | | | | |
| B5. Hypotension | Transient, intermittent, | Symptomatic, without | Syncope or symptomatic, | Shock |
| (without underlying | asymptomatic | interference with | interferes with function, | |
| diagnosis) | orthostatic decrease in | function, recurrent or | requiring therapy and | |
| | blood pressure> 20 mm | persistent > 20 mm Hg | sustained medical | |
| | Hg | decrease, responds to | attention, dose | |
| | | treatment | adjustment or drug | |
| | | | discontinuation | |
| B6. Myocardial | Transient chest | Recurring chest pain, | Angina with infarction, | Acute myocardial |
| ischaemia | pain/ECG changes; | transient ECG ST-T | no or minimal functional | infarction, arrhythmia |
| | rapid relief with nitro | changes; treatment | compromise, reduce dose | or/and CHF |
| | | relieves | or discontinue study drug | |
| B7. | Rub heard, | Detectable effusion by | Detectable on chest x- | Pulsus alternates with |
| Pericarditis/pericardial | asymptomatic | echocardiogram, | ray, dyspnea; or | low cardiac output; |
| effusion | | symptomatic, NSAID | pericardiocentesis; | requires surgery |
| | | required | requires corticosteroids | |
| B8. | Asymptomatic, | Symptomatic, recurrent, | Deep vein thrombosis | Pulmonary embolism |
| Phlebitis/thrombosis/ | superficial, transient, | deep vein thrombosis, no | requiring anticoagulant | |
| embolism (excludes | local, or no treatment | anticoagulant therapy | therapy | |
| injection sites) | required | required | | |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| C. GENERAL (constitutional) | tional) | | | |
| C1. Fatigue/malaise | Increase over baseline; | Limits daily function | Interferes with basic | Unable to care for self, |
| (asthenia) | most usual daily | intermittently over time | ADL, persistent | bed or wheelchair bound |
| | functions maintained, | | | > 50% of day |
| | short term | | | debilitating, |
| | | | | hospitalisation |
| C2. Fever (pyrexia) | Transient, few | Symptomatic, recurrent, | $\geq 40^{\circ}$ C; $\leq 24$ h, persistent | $\geq 40^{\circ}$ C, debilitating, |
| (note: fever due to | symptoms 37.7–38.5°C | 38.6-39.9°C. Relieved by | | > 24h, hospitalisation; no |
| drug allergy should be | | meds. | response to meds. | relief with meds |
| coded as allergy) | | | | |
| C3. Headache | Transient or | Persistent, recurring, | Prolonged, with limited | Intractable, debilitating, |
| | intermittent, no meds or | non-narcotic analgesics | response to narcotic | requires parenteral meds. |
| | relieved with OTC | relieve | medicine | |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life |
|---|---|---|---|---|
| C. GENERAL | | | | Till Catching |
| C4. Insomnia | Difficulty sleeping, | Difficulty sleeping, | Prolonged symptoms, | Debilitating, |
| | short term, not | interfering with function, | with limited response to | hospitalisation; no relief |
| | interfering with | use of prescription med. | narcotic meds. | with meds |
| | function | | | |
| C5. Rigors, chills | Asymptomatic, | Symptomatic, narcotic | Prolonged symptoms, | Debilitating, |
| | transient, no meds, or | meds relieve. | with limited response to | hospitalisation; no relief |
| | non-narcotic meds | | narcotic meds. | with meds |
| | relieve | | | |
| C6. Sweating | Episodic, transient | Frequent, short term | Frequent, drenching, | Dehydration, requiring |
| (diaphoresis) | | | disabling | IV fluids/hospitalization |
| | | | | > 24hr |
| C7. Weight gain | 5-9.9% | 10–19.9% | 20–30% | NA |
| C8. Weight loss | 5-9.9% | 10–19.9% | 20–30% | NA |

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| D. DERMATOLOGIC | | | | |
| D1. Alopecia | Subjective, transient | Objective, fully | Patchy, wig used, partly | Complete or irreversible |
| | | reversible | reversible | even if patchy |
| D2. Bullous eruption | Localised, | Localised, symptomatic, | Generalised, responsive | Prolonged, generalised, |
| | asymptomatic | requiring treatment | to treatment; reversible | or requiring |
| | | | | hospitalisation for |
| | | | | treatment |
| D3. Dry skin | Asymptomatic, | Symptoms eventually (1- | Generalised, interfering | Disabling for extended |
| | controlled with | 2 wks) controlled with | with ADL >2 wks, | period, unresponsive to |
| | emollients | emollients | persistent pruritus, | ancillary therapy and |
| | | | partially responsive to | requiring study drug |
| | | | treatment | discontinuation for relief |
| D4. Injection site | Local erythema, pain | Erythema, pain, oedema, | Prolonged induration, | Major ulceration necrosis |
| reaction | pruritus, < few days | may include superficial | superficial ulceration; | requiring surgery |
| | | phlebitis, 1-2 wks | includes thrombosis | |
| D5. Petechiae | Few, transient | Dependent areas, | Generalised, responsive | Prolonged, irreversible, |
| (without vasculitis) | asymptomatic | persistent up to 2 wks | to treatment; reversible | disabling |
0.: c02318676-08

Trial Protocol 

| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life |
|---|---|---|---|---|
| | | | | Hileatennig |
| D. DERMATOLOGIC | | | | |
| D6. Photosensitivity | Transient erythema | Painful erythema and | Blistering or | Generalised exfoliation |
| | | oedema requiring topical | desquamation, requires | or hospitalisation |
| | | treatment | systemic corticosteroids | |
| D7. Pruritus | Localised, | Intense, or generalised, | Intense or generalised; | Disabling, irreversible |
| | asymptomatic, | relieved by systematic | poorly controlled despite | |
| | transient, local | medication | treatment | |
| | treatment | | | |
| D8. Rash (not bullous) | Erythema, scattered | Diffuse macular/papular | Generalised, moist | Exfoliative or ulcerating; |
| | macular/papular | eruption or erythema | desquamation, requires | or requires |
| | eruption; pruritus | with pruritus; dry | systemic corticosteroids; | hospitalisation; or |
| | transient, OTC or no | desquamation; treatment | responsive to treatment; | parenteral corticosteroids |
| | meds | required | reversible | |
| D9. | Localized, high density | Local areas < 50% body | Generalised, disfiguring, | Disabling, irreversible, |
| Induration/fibrosis/ | on palpation, reversible, | surface, not disfiguring, | interferes with ADL, | systemic symptoms |
| Thickening (not | no effect on ADL and | transient interference | reversible | |
| sclerodermal) | no disfiguring | with ADL, reversible | | |
| scierodermai) | no distiguring | with ADL, reversible | | |

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| E. EAR/NOSE/THROAT | ΙΤ | | | |
| E1. Hearing loss | Transient, intermittent, | Symptomatic, treatment | Interferes with function; | Irreversible deafness |
| | no interference with | required, reversible | incomplete response to | |
| | function | | treatment | |
| E2. Sense of smell | Slightly altered | Markedly altered | Complete loss, reversible | Complete loss, without |
| | | | | recovery |
| E3. Stomatitis | Asymptomatic | Painful, multiple, can eat | Interferes with nutrition, | Requires enteral support, |
| | | | slowly reversible | residual dysfunction |
| E4. Taste disturbance | Transiently altered; | Persistently altered; | Disabling, effect on | NA |
| (dysgeusia) | metallic | limited effect on eating | nutrition | |
| E5. Tinnitus | Intermittent, transient, | Requires treatment, | Disabling, or associated | Irreversible deafness |
| | no interference with | reversible | with hearing loss | |
| | function | | | |
| E6. Voice changes | Intermittent hoarseness, | Persistent hoarseness, | Whispered speech, slow | Unable to vocalize for |
| (includes hoarseness, | able to vocalise | able to vocalise | return of ability to | extended |
| loss of voice, | | | vocalise | |
| laryngitis) | | | | |

Trial Protocol


| 4 - Includes Life<br>Threatening | | Extended duration | interference with | nutrition, requires | parenteral nutrition | | NA | | | | NA | | | | NA | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 3 - Severe | | Interferes with nutrition, | slowly reversible | | | | Symptoms impairing | function, vision loss | requiring treatment, | including surgery | ged, | partial response to | treatment, interferes with | function | Unresponsive to | treatment with major | effect on function |
| 2 - Moderate | | Relief with meds | | | | | Symptomatic, partial | visual loss, progressive | | | Symptomatic, responds | to treatment, changes not | interfering with function | | Symptomatic, treatment | required, reversible | |
| 1 - Mild | L | Transient dryness | | | | TOGIC | Asymptomatic, no | change in vision, non- | progressive | | Asymptomatic, | transient, rapid | response to treatment | | Symptoms not requiring Symptomatic, treatment | treatment, transient | |
| | E. EAR/NOSE/THROAT | E7. Xerostomia (dry | mouth) | | | F. EYE/OPHTHALMOLOGIC | F1. Cataract | | | | F2. Conjunctivitis | | | | F3. Lacrimation | increased (tearing, | watery eyes) |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| F. EYE/OPHTALMOLOGIC | OGIC | | | |
| F4. Retinopathy | Asymptomatic, non- | Reversible change in | Disabling change in | Loss of sight |
| | progressive, no | vision; readily responsive | vision ophthalmological | |
| | treatment | to treatment | findings reversible, sight | |
| | | | improves over time | |
| F5. Vision changes | Asymptomatic, | Symptomatic, vision | Symptomatic, vision | Loss of sight |
| (e.g. blurred, | transient, no treatment | changes not interfering | changes interfering with | |
| photophobia, night | required | with function, reversible | function | |
| blindness, vitreous | | | | |
| floaters) | | | | |
| F6. Xerophthalmia | Mild scratchiness | Symptomatic without | Interferes with | Loss of sight |
| (dry eyes) | | interfering with function, | vision/function, corneal | |
| | | requires artificial tears | ulceration | |
| G. GASTROINTESTINAL | IAL | | | |
| G1. Anorexia | Adequate food intake, | Symptoms requiring oral | Prolonged, requiring iv | Requires hospitalization |
| | minimal weight loss | nutritional | support | for nutritional support |
| | | supplementation | | |

: c02318676-08

Trial Protocol


| | | | | 0 |
|---|---|---|---|---|
| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life |
| | | | | Threatening |
| G. GASTROINTESTINAL | NAL | | | |
| G2. Constipation | Asymptomatic, | Symptomatic, requiring | Obstipation, requiring | Bowel obstruction. |
| | transient, responds to | prescription laxatives, | medical intervention | Surgery required. |
| | stool softener, OTC | reversible | | |
| | laxatives | | | |
| G3. Diarrhea | Transient, increase of | Symptomatic, increase | Increase > 6 stools/day, | Prolonged, dehydration, |
| | 2–3 stools/day over pre- | 4–6 stools/day, nocturnal | associated with disabling | unresponsive to |
| | treatment (no blood or | stools, cramping, | symptoms, e.g. | treatment, requires |
| | mucus), OTC agents | requires treatment with | incontinence, severe | hospitalization. |
| | relieve | prescription meds. | cramping, partial | |
| | | | response to treatment | |
| G4. Dyspepsia | Transient, intermittent, | Prolonged, recurrent, | Persistent despite | NA |
| (heartburn) | responds to OTC | requires prescription | treatment, interferes with | |
| | antacids, H-2 blockers | meds, relieved by meds | function, associated with | |
| | | | GI bleeding | |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| G. GASTROINTESTINAL | AL | | | |
| G5. GI bleed | Asymptomatic, | Symptomatic, transfusion | Haematemesis, | Recurrent, transfusion > |
| (gastritis, gastric or | endoscopic finding, | <pre>&lt;2 units needed;</pre> | transfusion 3–4 units, | 4 units, perforation, |
| duodenal ulcer | haemocult + stools, no | responds to treatment | prolonged interference | requiring surgery, |
| diagnosed-define | transfusion, responds | | with function | hospitalisation |
| aetiology) | rapidly to treatment | | | |
| G6. Haematochezia | Haemorrhoidal, | Symptomatic, transfusion | Recurrent, transfusion > | > 4 units, hypotension, |
| (rectal bleeding) | asymptomatic, no | <pre>&lt;2 units, reversible</pre> | 3–4 units | requiring hospitalization |
| | transfusion | | | |
| G7. Hepatitis | Laboratory | Symptomatic laboratory | Laboratory abnormalities | Progressive, hepato- |
| | abnormalities, | abnormalities, not | persistent >2wks, | renal, anasarca, pre-coma |
| | asymptomatic, | interfering with function, | symptoms interfere with | or coma |
| | reversible | slowly reversible | function | |
| G8. Nausea, or | Transient, intermittent, | Persistent, recurrent, | Prolonged, interferes | Hypotensive, |
| nausea/vomiting (use | minimal interference | requires prescription | with daily function and | hospitalization, |
| diagnostic term) | with intake, rapid | meds, intake maintained | nutritional intake, | parenteral nutrition, |
| | response to meds. | | periodic iv fluids | unresponsive to out- |
| | | | | patient management |


Bochringer Ingelheim BI Trial No.: 1311.13 Doc. No.: c02318676-08

c02318676-08 Trial Protocol

| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life |
|---|---|---|---|---|
| | | | | Threatening |
| G. GASTROINTESTINAL | VAL | | | |
| G9. Pancreatitis | Amylase elevation, | Amylase elevation with | Severe, persistent | Complicated by shock, |
| | intermittent | abdominal pain, nausea, | abdominal pain with | haemorrhage (acute |
| | nausea/vomiting, | occasional vomiting, | pancreatic enzyme | circulatory failure) |
| | transient, responds | responsive to treatment | elevation, incomplete or | |
| | rapidly to treatment | | slow response to | |
| | | | treatment | |
| G10. Proctitis | Perianal pruritus, | Tenesmus or ulcerations, | Unresponsive to | Mucosal necrosis with |
| | haemorrhoids (new | anal fissure, responsive | treatment, marked | haemorrhage, infection, |
| | onset), transient, or | to treatment, minimal | interference with | surgery required. |
| | intermittent, relieved by | interference with | function | |
| | OTC meds | function | | |
| H. MUSCULOSKELETAL | TAL | | | |
| H1. Avascular | Asymptomatic | MRI changes and | MRI changes, symptoms | Wheelchair bound; |
| necrosis | Magnetic resonance | symptoms responsive to | requiring surgical | surgical repair not |
| | imaging (MRI) | rest and analgesia | intervention | possible |
| | changes, non- | | | |
| | progressive | | | |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| H. MUSCULOSKELETAL | [AL] | | | |
| H2. Arthralgia | Intermittent transient symptoms, no meds or relieved by OTC meds | Persistent or recurrent symptoms, resolve with meds, little effect on | Severe symptoms despite<br>meds impairs function | Debilitating,<br>hospitalisation required<br>for treatment |
| H3. Leg cramps | Transient, intermittent, does not interfere with function | Recurrent symptoms, minimally interferes with function or sleep, respond to meds | Persistent, prolonged interference with function or sleep, partial or no response to meds | NA |
| H4. Myalgia | Occasional; does not interfere with function | Frequent, requires meds (non- narcotic); minor effect on function | Major change in function/lifestyle, narcotic pain meds | Debilitating, profound weakness, requires wheelchair, unresponsive to meds |
| I. NEUROPSYCHIATRIC | AC | | | |
| I-1. Anxiety or<br>Depression (mood<br>alteration) | Symptomatic, does not interfere with function; no meds | Frequent symptoms, responds to meds; interferes with ADL at times | Persistent, prolonged symptoms; partial or no response to meds, limits daily function | Suicidal ideation or danger to self |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.


Boehringer Ingelheim BI Trial No.: 1311.13

BI 1 rial No.: 1311.13 Doc. No.: c02318676-08

Trial Protocol

| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life |
|---|---|---|---|---|
| | | | | Threatening |
| I. NEUROPSYCHIATRIC | AC | | | |
| I-2. Cerebrovascular | NA | Single transient | Recurrent transient | Cerebrovascular vascular |
| ischaemia | | ischaemic event, | ischemic events | accident with permanent |
| | | responsive to treatment | | disability |
| I-3. Cognitive | Subjective symptoms, | Objective symptoms, | Persistent, or worsening | Debilitating/disabling |
| disturbance | transient, intermittent, | persisting, interferes with | objective symptoms; | and permanent; toxic |
| | not interfering with | daily function | interferes with daily | psychosis |
| | function | occasionally | routine | |
| I-4. Depressed | Observed, transient, | Somnolence or sedation, | Persistent, progressive, | Coma |
| consciousness | intermittent, not | interfering with function | obtundation, stupor | |
| (somnolence) | interfering with | | | |
| | function | | | |
| I-5. Inability to | Subjective symptoms, | Objective findings, | Persistent, prolonged | NA |
| concentrate | does not interfere with | interferes with function | objective findings; or | |
| | function | | organic cause | |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| I. NEUROPSYCHIATRIC | ac | | | |
| I-6. Insomnia (in | Occasional difficulty | Recurrent difficulty | Persistent or worsening | NA |
| absence of pain) | sleeping, transient | sleeping; requires meds | difficulty sleeping; | |
| | intermittent, not | for relief; occasional | severely interferes with | |
| | interfering with | interference with | routine daily function | |
| | function | function | | |
| I-7. Libido decreased | Decrease in interest | Loss of interest; | Persistent, prolonged, | NA |
| | | influences relationship | interfering with | |
| | | | relationship | |
| I-8. Peripheral motor | Subjective or transient | Objective weakness, | Objective weakness with | Paralysis |
| neuropathy | loss of deep tendon | persistent, no significant | substantial impairment of | |
| | reflexes; function | impairment of daily | function | |
| | maintained | function | | |
| I-9. Peripheral sensory | Subjective symptoms | Objective sensory loss, | Prolonged sensory loss or | NA |
| neuropathy (sensory | without objective | persistent, not interfering | paraesthesias interfering | |
| disturbance) | findings, transient, not | with function | with function | |
| | interfering with | | | |
| | function | | | |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Trial Protocol


| rence of old res, controlled with iment of medication stive findings, ent, meds relieve, ionally interfering unction zing, requires oral occasional erence with on stent, requires | | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life |
|---|---|---|---|---|---|
| Recurrence of old seizures, controlled with adjustment of medication adjustment of medication (b) cocasional wheeze, no interference with activities occasional OTC meds occasional OTC meds occasional occasional occasional occasional of the function occasional oc | T VIII OX ON ON I I III VI | (10 | | | Hileatennig |
| Recurrence of old seizures, controlled with adjustment of medication adjustment of medication (Subjective symptoms, transient, intermittent, no treatment occasionally interfering with function (Meezing, requires oral interference with activities (Interference with function (Interfe | I. NEUROPSYCHIAI K | ALC: | | | |
| seizures, controlled with adjustment of medication Subjective symptoms, transient, intermittent, occasionally interfering with function NARY Occasional wheeze, no interference with function Transient, intermittent, persistent, requires occasional OTC meds narcotic or other relieve | I-10. Seizure | NA | Recurrence of old | Recurrence/exacerbation | Recurrence not |
| Subjective symptoms, transient, intermittent, no treatment of medication with function with function interference with activities occasional OTC meds occasional of the function interference with function meds, occasional occasional of function relieve prescription meds for function relieve prescription meds for function relieve function functi | | | seizures, controlled with | with partial response to | controlled, requiring |
| Subjective symptoms, recurrent, meds relieve, no treatment occasionally interfering with function with recurrence or interference with function function activities relieve occasional OTC meds occasional or relieve relieve symptoms, occasional of the function relieve prescription meds for relieve ransient, intermittent, prescription meds for relieve relieve prescription meds for transient intermittent, prescription meds for relieve relieve resumble function received for the function received for the function received for function fun | | | adjustment of medication | medication | hospitalization; new |
| yo Subjective symptoms, Objective findings, transient, intermittent, necurrent, meds relieve, no treatment with function with function with received with needs, no interference with function activities function function function relieve prescription meds for relieve prescription meds for prescription meds for fransient, intermittent, prescription meds for relieve | | | | | seizures |
| VARY Occasional wheeze, no interference with activities Transient, intermittent, occasional meds relieve, with function with function Transient, intermittent, persistent, requires occasional OTC meds occasional OTC meds prescription meds for prescription meds for function func | I-11. Vertigo | Subjective symptoms, | Objective findings, | Persistent, prolonged, | Debilitating without |
| NARY Occasional wheeze, no interference with activities Transient, intermittent, occasional OTC meds occasional OTC meds relieve occasional OTC meds relieve occasional other occasional or function occasional occasional or function occasional or function occasional occ | (dizziness) | transient, intermittent, | recurrent, meds relieve, | interfering with daily | response to medication, |
| MARY Occasional wheeze, no interference with activities Transient, intermittent, Persistent, requires or occasional OTC meds relieve with function function function prescription meds for relieve | | no treatment | occasionally interfering | function; partial response | hospitalization |
| NARY Occasional wheeze, no interference with activities Transient, intermittent, occasional OTC meds occasional OTC meds prescription meds for relieve | | | with function | to medication | |
| Occasional wheeze, no Wheezing, requires oral interference with meds, occasional activities function Transient, intermittent, Persistent, requires occasional OTC meds narcotic or other relieve prescription meds for | J. PULMONARY | | | | |
| interference with meds, occasional activities interference with function Transient, intermittent, Persistent, requires occasional OTC meds narcotic or other relieve prescription meds for | J1. Asthma | Occasional wheeze, no | Wheezing, requires oral | Debilitating, requires | Requires ventilator |
| activities interference with function Transient, intermittent, Persistent, requires occasional OTC meds narcotic or other relieve prescription meds for | | interference with | meds, occasional | nasal $O_2$ | assistance |
| Transient, intermittent, Persistent, requires occasional OTC meds narcotic or other relieve prescription meds for | | activities | interference with | | |
| Transient, intermittent, Persistent, requires occasional OTC meds narcotic or other relieve prescription meds for | | | function | | |
| onal OTC meds narcotic or other prescription meds for | J2. Cough | | Persistent, requires | Recurrent, persistent | Interferes with |
| prescription meds for | | _ | narcotic or other | coughing spasms without | oxygenation; debilitating |
| | | relieve | prescription meds for | consistent relief by meds, | |
| | | | relief | interferes with function | |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| J. PULMONARY | | | | |
| J3. Dyspnea | Subjective, transient, no interference with function | Symptomatic, intermittent or recurring, interferes with exertional | Symptomatic during daily routine activities, interferes with function, | Symptomatic at rest, debilitating, requires constant nasal O <sub>2</sub> |
| | | activities | treatment with intermittent nasal O <sub>2</sub> relieves | |
| J4. Pleuritic pain (pleurisy) | Transient, intermittent symptoms, no treatment or OTC meds relieve | Persistent symptoms, requires prescription meds for relief | Prolonged symptoms,<br>interferes with function,<br>requires frequent narcotic<br>pain relief | Debilitating, requiring hospitalisation |
| J5. Pneumonitis<br>(pulmonary infiltrates) | Asymptomatic radiographic changes, transient, no treatment required | Symptomatic, persistent, requiring corticosteroids | Symptomatic, requiring treatment including O <sub>2</sub> | Debilitating, not reversible; or requiring assisted ventilation |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

Boehringer Ingelheim BI Trial No.: 1311.13

Doc. No.: c02318676-08

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| J. PULMONARY | | | | |
| J6. Pulmonary | -ead jo %06-9 <i>L</i> | 51–75% of pre-treatment | 51–75% of pre-treatment 26–50% of pre-treatment | <25% of pre-treatment |
| function decreased | treatment value | value | value | value |
| (Forced vital capacity | | | | |
| (FVC) or carbon | | | | |
| monoxide diffusion | | | | |
| capacity—DLCO) | | | | |
| LABORATORY DATA | 1 | | | |
| K. HAEMATOLOGY | | | | |
| K1. Hgb (g/dl) | 1.0–1.4 | 1.5–2.0 | 2.1-2.9; or Hgb $< 8.0$ , $>$ | $\geq 3.0$ ; or Hgb < 7.0 |
| decrease from pre- | | | 7.0 | |
| treatment | | | | |
| K2. Leukopenia (total | 3.0–3.9 | 2.0–2.9 | 1.0-1.9 | < 1.0 |
| WBC) x $1000$ | | | | |
| K3. Neutropenia (x | 1.5–1.9 | 1.0–1.4 | 0.5-0.9 | < 0.5 |
| 1000) | | | | |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|
| LABORATORY DATA | | | | |
| K. HAEMATOLOGY | | | | |
| K4. Lymphopenia (x 1.5–1.9 1000) | 1.5–1.9 | 1.0–1.4 | 0.5–0.9 | < 0.5 |
| K5. Platelets (x 1000) 75– Lower limit of normal (LLN) | 75– Lower limit of normal (LLN) | 50–74.9 | 20–49.9; platelet transfusion required | < 20; recurrent platelet transfusions |
| LABORATORY DATA | | | | |
| L. CHEMISTRY | | | | |
| L1. Hypercalcaemia<br>(mg/dl) | 1.1 x ULN-11.5 | 11.6–12.5 | 12.6–13.5; or symptoms present | >13.5; or associated coma |
| L2. Hyperglycaemia (mg/dl)<br>Fasting | 140–160 | 161–250 | 251–500 | >500, or associated with fasting ketoacidosis |

80-92

Trial Protocol


| LABORATORY DATA 6.0-6.4 6.5-7.0 or any ECG > 7.0 or any arrh change L. CHEMISTRY 6.0-6.4 6.5-7.0 or any ECG > 7.0 or any arrh change L3. Hyperkalaemia 0.9 x LLN-7.8 7.7-7.0 6.9-6.5; or associated change < 6.5, or occurre with symptoms L6. Hypoglycemia 55-64 (no symptoms) 40-54 (or symptoms) 30-39 (symptoms impair < 30, or coma function) L7. Hyponatraemia NA 125-129 120-124 < 120 L7. Hyponatraemia NA 3.0-3.4 2.5-2.9 < 2.5 (mg/dl) L8. Hypokalaemia NA 3.0-3.4 2.5-2.9 < 2.5 (mg/dl) L9. CPK (also if 1.2-1.9 x ULN 2.0-4.0 x ULN veakness but without or symptoms or polymyositis- disease) rhabdomyolysis | | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life<br>Threatening |
|---|---|---|---|---|---|
| 5.5–5.9 6.0–6.4 6.5–7.0 or any ECG change 0.9 x LLN–7.8 7.7–7.0 8.9–6.5; or associated with symptoms 30–3.9 (symptoms impair function) NA 1.25–129 NA 3.0–3.4 2.5–2.9 NA 1.2–1.9 x ULN 2.0–4.0 x ULN se) September 1.2–1.9 x ULN september 2.5–2.9 Symptoms symptoms signs or symptoms symptoms | LABORATORY DATA | | | | |
| 5.5–5.9 6.0–6.4 6.5–7.0 or any ECG change 0.9 x LLN–7.8 7.7–7.0 6.9–6.5; or associated with symptoms 55–64 (no symptoms) 40–54 (or symptoms 30–39 (symptoms impair function) NA 125–129 120–124 NA 3.0–3.4 2.5–2.9 NA 3.0–3.4 2.5–2.9 NA 3.0–3.4 2.5–2.9 NA 3.0–3.4 2.5–2.9 NA seakness but without life-threatening signs or symptoms | L. CHEMISTRY | | | | |
| Change Change | L3. Hyperkalaemia | 5.5–5.9 | 6.0–6.4 | 6.5–7.0 or any ECG | > 7.0 or any arrhythmia |
| 0.9 x LLN-7.8 7.7-7.0 6.9-6.5; or associated with symptoms 55-64 (no symptoms) 40-54 (or symptoms) 30-39 (symptoms impair function) NA 125-129 120-124 NA 3.0-3.4 2.5-2.9 NA 2.0-4.0 x ULN > 4.0 x ULN with weakness but without life-threatening signs or symptoms | (mg/dl) | | | change | |
| NA 2.0-4.0 x ULN Symptoms with symptoms impair function function 1.2-1.9 x ULN 2.0-4.0 x ULN life-threatening signs or symptoms separation symptoms symptoms with symptoms symptoms with symptoms sympt | L5. Hypocalcaemia | 0.9 x LLN-7.8 | 7.7–7.0 | 6.9–6.5; or associated | < 6.5, or occurrence of |
| 55–64 (no symptoms) 40–54 (or symptoms 30–39 (symptoms impair function) 125–129 120–124 120–124 120–124 120–124 120–134 1.2–1.9 x ULN 2.0–4.0 x ULN weakness but without life-threatening signs or symptoms 1.2–1.9 x ULN 2.0–4.0 x ULN weakness but without signs or symptoms 1.2–1.9 x ULN 2.0–4.0 x ULN weakness but without signs or symptoms 1.2–1.9 x ULN 2.0–4.0 x ULN weakness but without 1.2–1.9 x ULN 2.0–4.0 x ULN weakness but without 1.2–1.9 x ULN 2.0–4.0 x ULN weakness but without 1.2–1.9 x ULN 2.0–4.0 x ULN x veakness but without 1.2–1.9 x ULN | (mg/dl) | | | with symptoms | tetany |
| NA 125–129 120–124 120–124 NA 3.0–3.4 2.5–2.9 1.2–1.9 x ULN 2.0–4.0 x ULN | L6. Hypoglycemia | 55-64 (no symptoms) | 40–54 (or symptoms | 30–39 (symptoms impair | < 30, or coma |
| NA 3.0–3.4 1.2–1.9 x ULN 2.0–4.0 x ULN weakness but without life-threatening signs or symptoms | (mg/dl) | | present) | function) | |
| NA 3.0–3.4 2.5–2.9 1.2–1.9 x ULN 2.0–4.0 x ULN weakness but without life-threatening signs or symptoms | L7. Hyponatraemia | NA | 125–129 | 120–124 | < 120 |
| 1.2–1.9 x ULN | (mg/dl) | | | | |
| 1.2–1.9 x ULN 2.0–4.0 x ULN weakness but without life-threatening signs or symptoms | L8. Hypokalaemia | NA | 3.0-3.4 | 2.5–2.9 | < 2.5 |
| 1.2–1.9 x ULN 2.0–4.0 x ULN weakness but without life-threatening signs or symptoms | (mg/dl) | | | | |
| weakness but without life-threatening signs or symptoms | L9. CPK (also if | 1.2–1.9 x ULN | 2.0-4.0 x ULN | > 4.0 x ULN with | > 4.0 x ULN with signs |
| | polymyositis- disease) | | | weakness but without | or symptoms of |
| | | | | life-threatening signs or | rhabdomyolysis or life- |
| | | | | symptoms | threatening |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

30 January 2018

Boehringer Ingelheim BI Trial No.: 1311.13

Doc. No.: c02318676-08

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life |
|---|---|---|---|---|
| | | | | Threatening |
| LABORATORY DATA | 4 | | | |
| L. CHEMISTRY | | | | |
| L10.Serum uric acid | 1.2–1.6 x ULN | 1.7–2.9 x ULN | 3.0–5.0 x ULN or gout | NA |
| L11. Creatinine | 1.1–1.3 x ULN | 1.3–1.8 x ULN | 1.9–3.0 x ULN | > 3.0 x ULN |
| (mg/dl) | | | | |
| L12. SGOT (AST) | 1.2–1.5 x ULN | 1.6-3.0 x ULN | 3.1-8.0 x ULN | > 8.0 x ULN |
| L13. SGPT (ALT) | 1.2–1.5 x ULN | 1.6–3.0 x ULN | 3.0-8.0 x ULN | > 8.0 x ULN |
| L14. Alkaline | 1.1–2.0 x ULN | 1.6–3.0 x ULN | 3.0-5.0 x ULN | > 5.0 x ULN |
| phosphatase | | | | |
| L15. T. bilirubin | 1.1–1.4 x ULN | 1.5–1.9 x ULN | 2.0–3.0 x ULN | > 3.0 x ULN |
| L16. LDH | 1.3-2.4 x ULN | $2.5-5.0 \times ULN$ | $5.1-10 \times \text{ULN}$ | > 10 x ULN |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

Trial Protocol


| | 1 - Mild | 2 - Moderate | 3 - Severe | 4 - Includes Life |
|---|---|---|---|---|
| | | | | Threatening |
| LABORATORY DATA | _ | | | |
| M. URINALYSIS | | | | |
| M1. Haematuria | Micro only | Gross, no clots | Clots, transfusion < 2 | Transfusions required |
| | | | units | |
| M2. Proteinuria (per | 300-500 mg (tr/1+) | 501–1999 mg (2+) | 2-5.0 mg (3+) nephrotic | > 5.0 g (4+) anasarca |
| 24 h) | | | syndrome | |
| M3. WBC in urine | NA | NA | Indicating acute | Associated with |
| | | | interstitial nephritis | acuterenal failure |
| M4. Uric acid crystals | Present without | NA | With stones or symptoms | Causing renal outflow |
| | symptoms | | of stones (e.g. renal | obstruction and |
| | | | colic) | hospitalization |

Proprietary confidential information. © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

## 11. DESCRIPTION OF GLOBAL AMENDMENT(S)

| Number of global amendment | 1 |
|---|---|
| Date of CTP revision | 26 September 2014 |
| EudraCT number | 2014-001687-36 |
| BI Trial number | 1311.13 |
| BI Investigational Product(s) | BI 655066 |
| Title of protocol | An open label extension trial assessing the safety |
| Title of protocol | and efficacy of BI 655066 administered |
| | subcutaneously in patients with moderate to |
| | severe chronic plaque psoriasis. |
| | severe chrome piaque psoriasis. |
| To be implemented only often | |
| To be implemented only after | |
| approval of the | |
| IRB/IEC/Competent Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | |
| IRB/IEC/ Competent | |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | |
| Section to be changed | CLINICAL TRIAL PROTOCOL SYNOPSIS, |
| | Trial site(s) |
| Description of change | Change wording to 'Multicenter, multi national' |
| Rationale for change | Number of sites and countries will change during |
| | the trial conduct. |
| Section to be changed | CLINICAL TRIAL PROTOCOL SYNOPSIS, |
| | Objective(s) |
| D : (: 6.1 | · |
| Description of change | Change from 'Long term' to 'Additional' safety |
| | and efficacy data. |
| Rationale for change | Modification of Objective to correlate with FDA |
| | requirement of maximum duration of |
| | administration of BI655066 of one year. |

| Section to be changed | CLINICAL TRIAL PROTOCOL SYNOPSIS, Duration of treatment |
|---|---|
| Description of change | Change from 'Approximately 4 years' to 'Maximum duration of administration to patient is one calendar year after receiving first dose of BI 655066' |
| Rationale for change | Modification to correlate with FDA requirement |
| Section to be changed | CLINICAL TRIAL PROTOCOL SYNOPSIS, Criteria for efficacy |
| Description of change | Modification of endpoint due to reduction in study duration and maximum administration of study medication of one year. |
| Rationale for change | Modification to correlate with FDA requirement |
| Section to be changed | FLOW CHART 1 |
| Description of change | Change of duration of treatment period and Follow up period, as well as correct footnotes and numbering. Additional text is added to footnote 1 to better explain roll-over from trial 1311.2, footnote 4 covering visits beyond visit 18 is deleted and wording for footnote 5 describing variable timing of EOT is modified to adapt the maximum duration of administration of one year. Corrective words have been added to footnote 9 and 12, Vital signs has been added to all scheduled visits, and footnote 19 has been added to better describe drug administration. |
| Rationale for change | These are administrative changes to correct duration of treatment period and follow up period, numbering of footnotes and to correct wordings in the footnotes to correlate with FDA requirement of maximum duration of administration of BI655066 of one year. |
| Section to be changed | 2.1 RATIONALE FOR PERFORMING THE TRIAL |
| Description of change | Change of wording from 'Long term' to 'Additional' safety and efficacy data, and add wording for 48 week follow up. |
| Rationale for change | Modification due to reduction in study duration and maximum administration of study medication of one year. |

| Section to be changed Description of change | 2.2 TRIAL OBJECTIVES |
|---|---|
| Description of change | Change of wording from 'Long term' to |
| • | 'Additional' safety and efficacy data. |
| Rationale for change | Modification due to reduction in study duration to |
| Rationale for change | one year administration of study medication. |
| | one year administration of study medication. |
| Section to be changed | 2.3 BENEFIT – RISK ASSESSMENT |
| Description of change | Further description of signs of hypersensitive |
| | reactions is added. |
| Rationale for change | Include further, adequate details concerning the |
| | performance of monitoring after IMPs injections, |
| | for all treated patients. |
| Section to be changed | 3.1 OVERALL TRIAL DESIGN AND PLAN |
| Section to be changed Description of change | Change of wording from 'Long term' to |
| Description of change | 'Additional' safety and efficacy data. |
| Rationale for change | · |
| Rationale for change | • |
| | one year administration of study medication. |
| Section to be changed | 3.1 OVERALL TRIAL DESIGN AND PLAN |
| Description of change | Description of how to proceed if a subject is |
| | eligible for 1311.13 and the protocol is not yet |
| | approved. |
| Rationale for change | |
| | specified. |
| Section to be changed | 3.1 OVERALL TRIAL DESIGN AND PLAN |
| 2 contiputed of change | |
| Rationale for change | |
| 8- | different visit throughout the trail. |
| Section to be changed | 3.1 OVERALL TRIAL DESIGN AND PLAN |
| - and promote than go | |
| Rationale for change | |
| | applicable in this trial. |
| Description of change | Description of how to proceed if a subject is eligible for 1311.13 and the protocol is not yet approved. To be able to re-evaluate subjects eligible for 1311.13 while protocol not yet approved. This situation is applicable for possible roll-overs from 1311.2 during the period the study initiation has been on hold. Procedures for re-evaluation is specified. 3.1 OVERALL TRIAL DESIGN AND PLAN Figure 3.1:2 'Drug Administration in trial 1311.13' is added Table is added to explain drug administration at different visit throughout the trail. 3.1 OVERALL TRIAL DESIGN AND PLAN Delete text describing adjustment of dosing to 180 mg and text describing possible reduction of dosing after study data from 1311.2 is revealed. Due to FDA regulation, maximum dosage is 90 mg per 12 week, 180 mg dose is no longer |

| Section to be changed | 3.1 OVERALL TRIAL DESIGN AND PLAN |
|---|---|
| Description of change | PASI <sub>75</sub> is added as standard clinical endpoint and |
| | to be assessed at each visit. |
| Rationale for change | The plaque psoriasis will be evaluated by PASI |
| | score at each visit. The standard clinical endpoints |
| | of PASI <sub>50</sub> , PASI <sub>75</sub> and PASI <sub>90</sub> will be assessed at |
| | each visit. |
| | TYG 2 1 2 G 11 11 G |
| Section to be changed | FIG 3.1:2 Guideline for assessment dose |
| | adjustment |
| Description of change | Figure is deleted. |
| Rationale for change | Figure describes possible dose adjustment |
| | between 90 mg and 180 mg dose. Due to FDA |
| | regulation, maximum dosage is 90 mg per 12 |
| | week, 180 mg dose is no longer applicable in this |
| | trial. |
| C-44-11 | 2.1.1 ADMINISTD ATIME STRUCTURE OF |
| Section to be changed | 3.1.1 ADMINISTRATIVE STRUCTURE OF |
| D | THE TRIAL |
| Description of change | Change of number of participating sites and |
| | countries. |
| Rationale for change | Number of participating sites and countries has |
| | been modified, to reflect the current status for |
| | this. |
| Section to be changed | 3.2 DISCUSSION OF TRIAL DESIGN |
| Description of change | Delete text describing adjustment of dosing to |
| Description of change | 180 mg. |
| Rationale for change | Due to FDA regulation, maximum dosage is 90 |
| reationale for change | mg per 12 week, 180 mg dose is no longer |
| | applicable in this trial. |
| | application in this trial. |
| Section to be changed | 3.2 DISCUSSION OF TRIAL DESIGN |
| <b>Description of change</b> | Change of wording from 'Long term' to |
| | 'Additional' safety and efficacy data, and adding |
| | 'following one year drug administration'. |
| Rationale for change | Modification due to reduction in study duration |
| | and administration of study medication. |
| | • |
| Section to be changed | 3.3.4.1 REMOVAL OF INDIVIDUAL |
| | PATIENTS |
| Description of change | Corrections to reflect new study duration of 48 |
| | week follow up instead of 15 days. |
| Rationale for change | Study duration changed to 48w follow up after |
| | one year maximum study drug administration. |

| Section to be changed | 4.1.2 METHOD OF ASSIGNING PATIENTS TO TREATMENT GROUPS |
|---|---|
| Description of shapes | Delete text describing adjustment of dosing to |
| Description of change | 180 mg. |
| Dationals for shange | Due to FDA regulation, maximum dosage is 90 |
| Rationale for change | mg per 12 week, 180 mg dose is no longer |
| | applicable in this trial. |
| | applicable in this trial. |
| Section to be changed | 4.1.3 SELECTION OF DOSES IN THE TRIAL |
| Description of change | Delete text describing adjustment of dosing to |
| | 180 mg and possible adjustment of dosing once |
| | the 1311.2 study results are available. |
| Rationale for change | Due to FDA regulation, maximum dosage is 90 |
| | mg per 12 week, 180 mg dose is no longer |
| | applicable in this trial.dose applicable for this |
| | study. |
| G. A. L. L. L. L. | TADLE 41.41 Days was in an |
| Section to be changed | TABLE 4.1.4.1. Dose regimens |
| Description of change | Table is deleted. |
| Rationale for change | Table describes dose regimens for 90 mg and 180 |
| | mg dose. Dose of 90 mg is the only dose |
| | applicable for this study. |
| Section to be changed | 4.1.4 DOSE ASSIGNMENT AND |
| | ADMINISTRATION OF DOSES |
| Description of change | Further description of signs of hypersensitive |
| | reactions is added. |
| Rationale for change | Include further, adequate details concerning the |
| | performance of monitoring after IMPs injections, |
| | for all treated patients. Requirement from French |
| | HA. |
| Section to be changed | 5.1.1 ENDPOINTS OF EFFICACY |
| Description of change | Time of evaluation of primary and secondary |
| Description of change | endpoints has been changed from 12 week to 48 |
| | week. |
| Rationale for change | Change of timing of evaluation for endpoints |
| Rationale for change | necessary to reflect maximum study drug |
| | administration of one calendar year. |
| | administration of one calcular year. |

| Section to be changed | TABLE 5.2.3:2 SAFETY LABORATORY<br>TESTS |
|---|---|
| Description of change | Test for ESR (erythrocyte sedimentation rate after 1 hour) is deleted. |
| Rationale for change | ESR test is not to be performed, due to evaluations from 1311.2. The test had to be performed at local lab, and the interpretation of the test results is not validated to give reliable values. |
| Section to be changed | 6.2.2 TREATMENT PERIOD(S) |
| Description of change | Description of how to proceed if a subject is eligible for 1311.13 and the amended protocol is not yet approved. Also added in section 3.1. |
| Rationale for change | To be able to re-evaluate subjects eligible for 1311.13 while protocol not yet approved. This situation is applicable for possible roll-overs from trial 1311.2 during the period the study 1311.13 has not yet been initiated due to review of protocol amendment. Procedures for re-evaluation are specified. |
| Section to be changed | 6.2.2 TREATMENT PERIOD(S) |
| Description of change | Text describing adjustment of dosing to 180 mg is deleted. |
| Rationale for change | Dose of 90 mg is the only dose applicable for this study. |
| Section to be changed | 6.2.3 END OF TRIAL AND FOLLOW_UP<br>PERIOD |
| Description of change | Specification of end of trial is changed, adding description of 48 week follow up period. |
| Rationale for change | Specification of end of trial is changed due to reduction in study duration and administration of study medication of maximum one year. |
| Section to be changed | 7.2 NULL AND ALTERNATIVE HYPETHESIS |
| Description of change | Change of wording regarding duration of study drug administration. |
| Rationale for change | Modification due to reduction in study duration and maximum administration of study medication of one year. |

| Section to be changed | 7.3 PLANNED ANALYSIS |
|-----------------------|-------------------------------------------------|
| Description of change | Deleting text describing critical time-points |
| | beyond 1 year. |
| Rationale for change | Modification due to reduction in study duration |
| | and maximum administration of study medication |
| | of one year. |
| Section to be changed | 7.3.1 PRIMARY ANALYSIS |
| Description of change | Modification of endpoint due to reduction in |
| | study duration and maximum administration of |
| | study medication of one year. |
| Rationale for change | Modification to correlate with FDA requirement |

| Number of global amendment | 2 |
|---|---|
| Date of CTP revision | 15 October 2014 |
| EudraCT number | 2014-001687-36 |
| BI Trial number | 1311.13 |
| BI Investigational Product(s) | BI 655066 |
| Title of protocol | An open label extension trial assessing the safety and efficacy of BI 655066 administered subcutaneously in patients with moderate to severe chronic plaque psoriasis. |
| To be implemented only often | |
| To be implemented only after | |
| approval of the | |
| IRB/IEC/Competent | |
| Authorities To be implemented | |
| To be implemented immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | |
| IRB/IEC/ Competent | |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | |
| Section to be changed | FLOW CHART 1 |
| Description of change | Change of wording for day and week to relate to EOT instead of absolute numbers. Change of text in footnote 4 to better explain drug administrations. Addition of footnote 20 and 21 to better explain procedures for prematurely discontinuation and collection of vital signs and vital status follow up. Assessment for Tolerability (safety and efficacy) has been deleted, as this was primarily for evaluation of dose adjustments which are no longer applicable, so has local |
| | tolerability test for follow up period after FU2. |
| Rationale for change | These are administrative changes to clarify timing of visit, and study procedures for drug administrations, withdrawals and collection of vital signs and vital status follow up. |

| Castina to be about | 2.1 OVED ALL TRIAL DECICN AND DUAN |
|---|---|
| Section to be changed | 3.1 OVERALL TRIAL DESIGN AND PLAN |
| Description of change | Study number 1311.13 added in text to clarify |
| | drug administration for patients that did not |
| | receive BI655066 in trial 1311.2 |
| Rationale for change | Text added to clarify. |
| Section to be changed | 3.1 OVERALL TRIAL DESIGN AND PLAN |
| Description of change | Figure 3.1:2 deleted and replaced by Flow Chart 2 |
| Description of change | to better explain drug administration |
| Rationale for change | Figure revised to clarify drug administration. |
| Kationale for Change | riguic levised to clarify drug administration. |
| Section to be changed | 3.3.4 REMOVAL OF PATIENTS |
| Description of change | Text added to clarify procedures for withdrawal |
| | in follow up period |
| Rationale for change | Text added to clarify. |
| Section to be changed | 5.2.5 ASSESSMENT OF OTHER SAFETY |
| | PARAMETER |
| Description of change | Text explaining 'Tolerability (safety and |
| | efficacy)' has been deleted, as this was primarily |
| | for evaluation of dose adjustments which are no |
| | longer applicable. |
| Rationale for change | Assessment no longer applicable, as only one |
| | dose applicable in this trial. |
| Section to be abanged | 6.2.2.TREATMENT PERIOD |
| Section to be changed | 'EOT' removed from text to avoid mix with EOS. |
| Description of change | |
| | Added text regarding study window removed, misleading. |
| Detienals for alcono | |
| Rationale for change | Text removed to clarify. |
| Section to be changed | 6.2.2.TREATMENT PERIOD |
| <b>Description of change</b> | Text added to clarify drug administration for |
| | patients that did not receive BI655066 in trial |
| | 1311.2. Also ref to Flow Chart 2 added to clarify. |
| Rationale for change | Text and reference to Flow Chart 2 added to |
| | clarify. |
| Section to be changed | 6.2.3 END OF TRIAL AND FOLLOW-UP |
| | PERIOD |
| Description of change | Text added to clarify procedures for withdrawal |
| | in follow up period |
| Rationale for change | Text added to clarify. |
| | CAA END OF EDITE AND FOLLOWING |
| Section to be changed | 6.2.3 END OF TRIAL AND FOLLOW-UP |
| Section to be changed Description of change | 6.2.3 END OF TRIAL AND FOLLOW-UP PERIOD Text added to describe collection of consent for |

## Proprietary confidential information.

| | vital status follow up. |
|---|---|
| Rationale for change | Text added to clarify. |
| Normalism of all hall are an illustrated | 3 |
| Number of global amendment Date of CTP revision | 10 June 2015 |
| EudraCT number | 2014-001687-36 |
| BI Trial number | 1311.13 |
| BI Investigational Product(s) | BI 655066 |
| Title of protocol | An open label extension trial assessing the safety |
| | and efficacy of BI 655066 administered |
| | subcutaneously in patients with moderate to |
| | severe chronic plaque psoriasis. |
| To be implemented only after | |
| approval of the | |
| IRB/IEC/Competent | |
| Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | |
| IRB/IEC/ Competent | |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | |
| Section to be changed | CLINICAL TRIAL PROTOCOL SYNOPSIS, |
| D : ( C) | Objective(s) |
| Description of change | Change from 'Additional' to 'Long term' safety |
| D. C. L. C. L. | and efficacy data. |
| Rationale for change | Return to original CTP wording with approx 4 |
| | years duration of treatment. New toxicity data |
| | cancel FDA requirement of maximum duration of |
| | administration of BI655066 of one year. |
| Section to be changed | CLINICAL TRIAL PROTOCOL SYNOPSIS, |
| | No. patients each treatment |
| <b>Description of change</b> | Text including possible increase to 180 mg dosing |
| | every 12 week is added. |
| Rationale for change | Possibility to increase to 180 mg dosing |
| | depending on efficacy at 12 week added Patients |

| | should all reach >PASI <sub>90</sub> . |
|---|---|
| | Should all leach /PAS190. |
| Section to be changed | CLINICAL TRIAL PROTOCOL SYNOPSIS,<br>Test product (s) |
| Description of change | '180 mg dosing every 12 week' added |
| Rationale for change | Possible increase to 180 mg dosing depending on efficacy at 12 week. |
| Section to be changed | CLINICAL TRIAL PROTOCOL SYNOPSIS, Duration of treatment |
| Description of change | Change from 'Maximum duration of one calendar year' to 'Approximately four years of administration'. '48 week follow up period' deleted. |
| Rationale for change | Return to original CTP wording with approx 4 years duration of treatment. New toxicity data cancel FDA requirement of maximum duration of administration of BI655066 of one year. Follow up period will now be REP i.e. 12 weeks. |
| Section to be changed | CLINICAL TRIAL PROTOCOL SYNOPSIS,<br>Criteria for efficacy |
| Description of change | Added 'in the Extended dosing period' |
| Rationale for change | To clarify that point of achievement will be at 48 week in the extended dosing period only. |
| Section to be changed | FLOW CHART |
| Description of change | Previous Flow Chart 1 deleted and replaced by a new. Visit scheduling of previous Flow Chart 1 is now added as Figure 3.1.3. New Flow Chart is called 'Extended dosing period'. Change of wording for visit to relate to Extended period. Footnotes added or modified to explain new study procedures related to the extension of the trial and possible re-start of treatment. |
| Rationale for change | Flow Chart has been modified to reflect procedures and timing related to the extension of the trial and possible re-start of treatment for the patients with low response ( <pasi<sub>90) at week 12.</pasi<sub> |
| Section to be changed | FLOW CHART 2 |
| Description of change | Flow Chart 2 is deleted. (Replaced by Fig 3.1.3) |
| Rationale for change | Flow Chart 2 is no longer applicable, due to no limitation of maximum one year dosing per |

| 1 | patient. Headings kept as reference in Fig 3.1.3 |
|---|---|
| | ADDREVIATIONS |
| Section to be changed Description of change | ABBREVIATIONS Abbreviations added for PASE, EV, OPU, ISF, |
| Description of change | Th and IgG. |
| Rationale for change | Missed or added since previous amendment. |
| Rationale for change | wissed of added since previous amendment. |
| Section to be changed | 2.1 RATIONALE FOR PERFORMING THE |
| | TRIAL |
| Description of change | Change from 'one' to 'approximately four years' |
| | treatment, '48 weeks follow up' deleted. |
| Rationale for change | Return to original CTP wording with approx 4 |
| | years duration of treatment. New toxicity data |
| | cancel FDA requirement of maximum duration of administration of BI655066 of one year. |
| | administration of Bio33000 of one year. |
| Section to be changed | 2.2 TRIAL OBJECTIVES |
| Description of change | Change from 'one' to 'approximately four years' |
| | treatment, change from 'up to one year' and |
| | 'additional' to 'long term'. |
| Rationale for change | Return to original CTP wording with approx 4 |
| | years duration of treatment. New toxicity data |
| | cancel FDA requirement of maximum duration of |
| | administration of BI655066 of one year. |
| Section to be changed | 2.3 BENEFIT – RISK ASSESSMENT |
| Section to be changed Description of change | 2.3 BENEFIT – RISK ASSESSMENT 'Visit 1' replaced by 'rollover visit' . 'Extended' |
| · | |
| | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial roll- |
| Description of change | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous |
| Description of change | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial roll- |
| Description of change | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. |
| Description of change Rationale for change Section to be changed | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN |
| Description of change Rationale for change | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four |
| Description of change Rationale for change Section to be changed Description of change | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four years' treatment. Description of study end added. |
| Description of change Rationale for change Section to be changed | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four years' treatment. Description of study end added. Return to original CTP wording with approx 4 |
| Description of change Rationale for change Section to be changed Description of change | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four years' treatment. Description of study end added. Return to original CTP wording with approx 4 years duration of treatment. The study is planned |
| Description of change Rationale for change Section to be changed Description of change | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four years' treatment. Description of study end added. Return to original CTP wording with approx 4 years duration of treatment. The study is planned to continue until marketing approval of BI655066 |
| Description of change Rationale for change Section to be changed Description of change | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four years' treatment. Description of study end added. Return to original CTP wording with approx 4 years duration of treatment. The study is planned |
| Description of change Rationale for change Section to be changed Description of change | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four years' treatment. Description of study end added. Return to original CTP wording with approx 4 years duration of treatment. The study is planned to continue until marketing approval of BI655066 |
| Description of change Rationale for change Section to be changed Description of change Rationale for change | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four years' treatment. Description of study end added. Return to original CTP wording with approx 4 years duration of treatment. The study is planned to continue until marketing approval of BI655066 in each country. |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four years' treatment. Description of study end added. Return to original CTP wording with approx 4 years duration of treatment. The study is planned to continue until marketing approval of BI655066 in each country. 3.1 OVERALL TRIAL DESIGN AND PLAN |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four years' treatment. Description of study end added. Return to original CTP wording with approx 4 years duration of treatment. The study is planned to continue until marketing approval of BI655066 in each country. 3.1 OVERALL TRIAL DESIGN AND PLAN Procedure for roll-over to 'Extended visit 1' |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four years' treatment. Description of study end added. Return to original CTP wording with approx 4 years duration of treatment. The study is planned to continue until marketing approval of BI655066 in each country. 3.1 OVERALL TRIAL DESIGN AND PLAN Procedure for roll-over to 'Extended visit 1' described in the text and Figure 3.2.3.added to refer to previous visit schedule. New visit schedule for 'Extended dosing period' |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed Description of change | 'Visit 1' replaced by 'rollover visit' . 'Extended' added. TB testing only to be performed at the initial rollover visit. Extended EOT replacing previous EOT. 3.1 OVERALL TRIAL DESIGN AND PLAN Change from 'total of one' to 'approximately four years' treatment. Description of study end added. Return to original CTP wording with approx 4 years duration of treatment. The study is planned to continue until marketing approval of BI655066 in each country. 3.1 OVERALL TRIAL DESIGN AND PLAN Procedure for roll-over to 'Extended visit 1' described in the text and Figure 3.2.3.added to refer to previous visit schedule. |


| | A 1 OVER ALL TRULL DEGICAL AND BUANT |
|---|---|
| Section to be changed | 3.1 OVERALL TRIAL DESIGN AND PLAN |
| Description of change | Figure 3.1.2.added |
| Rationale for change | Figure added to give guideline for assessment of |
| | dose adjustment. |
| Section to be changed | 3.1 OVERALL TRIAL DESIGN AND PLAN |
| Description of change | Figure 3.1.3.added |
| Rationale for change | Headings from previous Flow Chart kept as |
| Rationale for change | reference to visit schedule naming. |
| | reference to visit senedule naming. |
| | 2.1 OVER ALL TRIAL DEGICNI AND BLAN |
| Section to be changed | 3.1 OVERALL TRIAL DESIGN AND PLAN |
| Description of change | 'PASI <sub>100</sub> ' and 'Extended' added. |
| Rationale for change | To be in accordance with section 5.1.1.1.2 and |
| | 7.3.2. |
| Section to be changed | 3.1 OVERALL TRIAL DESIGN AND PLAN |
| Description of change | Number of sites and countries corrected. |
| Rationale for change | Since last AM, number of participating sites and |
| Rationale for change | countries has been modified. |
| | countries has been mouried. |
| Section to be changed | 3.2 DISUSION OF TRIAL DESIGN |
| Description of change | "option of moving to a higher dose (180 mg) if |
| | loss of clinically activity is noted' is added. |
| Rationale for change | Possible increase to 180 mg dosing depending on |
| | efficacy at 12 week. Patients should all reach |
| | >PASI <sub>90</sub> . |
| | A A GEV E CEVON OF EDIAN DODAY A EVON |
| Section to be changed | 3.3 SELECTION OF TRIAL POPULATION |
| Description of change | 'Visit 1' changed to 'roll-over visit' in inclusion |
| | and exclusion criteria. REP changed from 15 to |
| | 12 weeks. |
| Rationale for change | To adapt wording to new visit schedule naming |
| | and design. REP changed according to new IB ver |
| | 5 for BI 6550066. |
| Section to be changed | 3.3.4 REMOVAL OF PATIENTS FROM |
| | THERAPY |
| Description of change | Sentence regarding FU visit is deleted. |
| | 'Extended' added to all visits mentioned in the |
| | text. Follow up period changed from 48 to 12 |
| | weeks. 'Visit 1' replaced by 'roll-over visit'. |
| Rationale for change | FU visits no longer in the revised Flow Chart. |
| | 'Extended' added to reflect visit schedule naming |
| | in new flow Chart. |
| Section to be changed | 4.1 TREATMENT TO BE ADMINISTERED |
| | 4 1 1 1 1 1 2 4 1 1 1 1 1 1 1 1 1 |

| Description of change Rationale for change | Text added to describe possible increase in dosing to 180 mg if lack of response. Text to explain selection of dose has been modified. Instruction for injection of 180 mg added. Possible increase to 180 mg dosing depending on efficacy at 12 week. Text to explain selection of dose has been modified to reflect new findings |
|---|---|
| | from the interim analysis of 1311.2. |
| Section to be changed | 4.2.2 RESTRICTIONS |
| Description of change | 'Extended' added and Visit 1' changed to 'roll- |
| Description of change | over visit' in Table 4.2.2.1 |
| Rationale for change | 'Extended' added to reflect visit schedule naming in new flow Chart. |
| Section to be changed | 5.1 EFFICACY -PHARMACODYNAMICS |
| <b>Description of change</b> | 'in Extended dosing period' added in text. |
| Rationale for change | Added to clarify that prim endpoint will be achieved at 48 w in Extended dosing period only. |
| | demoted at 10 W in Entended dooring period omy. |
| Section to be changed | 5.2.2. ASSESSMENT OF ADVERSE EVENTS |
| Description of change | Time window for EV1 changed to 6 weeks. REP |
| | changed from 15 to 12 weeks. |
| Rationale for change | Time window for entering EV1 from EOS of 1311.2 changed from 7 days to 6 weeks, to be able to include patients that had to wait for the approval of this amendment for their roll-over. REP changed to 12 weeks/ 84 days according to IB ver 6 for IB655066. |
| Section to be changed | 5.2.3 ASSESSMENT OF SAFETY |
| D | LABORATORY PARAMETERS |
| Description of change | 'Visit 1' changed to 'roll-over visit' in table 5.2.3:2. 'Extended' added. |
| Rationale for change | Changed to clarify and reflect visit schedule |
| | naming in new flow Chart. |
| Section to be changed | 5.2.4 ELECTROCARDIOGRAM |
| Description of change | Specification of visits were ECG will be obtained |
| Description of change | is deleted. |
| Rationale for change | ECG will be obtained every 24 weeks according |
| | to new Flow Chart. |
| Section to be changed | 5.2.5 ASSESSMENT OF OTHER SAFETY |
| | PARAMETERS |
| <b>Description of change</b> | 'Visit 1' changed to 'roll-over visit' |
| Rationale for change | Changed to clarify procedure according to new visit schedule. |


| Section to be changed | 6.2.2 TREATMENT PERIOD |
|-----------------------|----------------------------------------------------|
| Description of change | Text modified and added to reflect procedures |
| | and assessments according to current Flow Chart. |
| Rationale for change | Flow Chart with footnotes covering Extended |
| | Dosing Period will replace former visit schedule |
| | and procedures. |
| Section to be changed | 6.2.3. END OF TRIAL AND FOLLOW UP |
| | PERIOD |
| Description of change | Text modified and added to reflect procedures |
| | and assessments according to current Flow Chart. |
| | Text regarding collection of vital status changed |
| | to open for collection of consent also at EV1. |
| Rationale for change | Flow Chart with footnotes covering Extended |
| | Dosing Period will replace former visit schedule |
| | and procedures. |
| Cooking to be about d | 7.1 STATISTICAL DESIGN |
| Section to be changed | |
| Description of change | Text 'single' arm replaced by 'double' arm. |
| Rationale for change | Double arm design due to introduction of possible |
| | 180 mg dose at EV2. |
| Section to be changed | 7.2 NULL AND ALTERNATIVE HYPETHESIS |
| Description of change | 'one year' replaced by 'extended visit period'. |
| Rationale for change | Text changed to reflect current visit schedule. |
| Section to be changed | 7.3 PLANNED ANALYSIS |
| Description of change | 'in Extended dosing period' added. REP changed |
| | to 12 weeks from 15 weeks. |
| Rationale for change | Added to specify time of efficacy endpoint. REP |
| | changed according to current IB ver 6. |
| Section to be changed | 10.5 PASE |
| Description of change | 'Visit 1' replaced by 'roll-over visit' to reflect |
| Description of change | current flow chart and procedures |
| Rationale for change | To reflect current flow chart and procedures for |
| Tanonaic ioi change | EV1. |

| | Τ |
|---|---|
| Number of global amendment | 4 |
| Date of CTP revision | 12 October 2016 |
| EudraCT number | 2014-001687-36 |
| BI Trial number | 1311.13 |
| BI Investigational Product(s) | BI 655066 |
| Title of protocol | An open label extension trial assessing the safety and efficacy of BI 655066/ ABBV-066/ (risankizumab) administered subcutaneously in patients with moderate to severe chronic plaque psoriasis. |
| To be implemented only after approval of the IRB/IEC/Competent Authorities | |
| To be implemented immediately in order to eliminate hazard – IRB / IEC / Competent Authority to be notified of change with request for approval | |
| Can be implemented without IRB/IEC/ Competent Authority approval as changes involve logistical or administrative aspects only | |
| | mid o |
| Section to be changed | Title page, Synopsis |
| Description of change | Changed BI drug or BI investigational product or BI 655066 to refer to either names for this compound: BI 655066/ ABBV-066/risankizumab. |
| Rationale for change | In February 2016, AbbVie entered into a license agreement with BI related to risankizumab, and in October 2016, the US IND for risankizumab transitioned from BI to AbbVie. This protocol change reflects that AbbVie will now be the Sponsor of this study in the US, as well as the modifications to certain study conduct responsibilities as a result of that license agreement are listed as separate changes below. |
| Section to be changed | 3.1.1 ADMINISTRATIVE STRUCTURE OF |
| Section to be changed | THE TDIAL |

Trial Protocol


| Description of change | <ol> <li>Changed sponsor from Boehringer Ingelheim (BI) to AbbVie in the US and BI for all other participating countries. </li> <li>Changed text to specify Statistical Evaluation</li> </ol> |
|---|---|
| | will be done by AbbVie according to their SOPs. |
| Rationale for change | Refer to rational for first change listed |
| Section to be changed | 3.3.4.2 DISCONTINUATION OF THE TRIAL |
| | BY THE SPONSOR |
| Description of change | Updated text to "AbbVie/Boehringer Ingelheim reserves the right to discontinue the trial overall or at a particular trial site at any time for the |
| | following reasons". |
| Rationale for change | Refer to rational for first change listed |

| Number of global amendment | 5 |
|---|---|
| Date of CTP revision | 30 January 2018 |
| EudraCT number | 2014-001687-36 |
| BI Trial number | 1311.13 |
| BI Investigational Product(s) | BI 655066 |
| Title of protocol | An open label extension trial assessing the safety and efficacy of BI 655066/ ABBV-066/ (risankizumab) administered subcutaneously in patients with moderate to severe chronic plaque psoriasis. |
| To be implemented only after | |
| approval of the | |
| IRB/IEC/Competent | |
| Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | |
| IRB/IEC/ Competent | |
| Authority approval as changes | |
| involve logistical or | |
| administrative aspects only | |
| Section to be changed | FLOW CHART-extended dosing period |
| Description of change | Added at the EOS visit: |
| r · | After the approval of this protocol amendment in |
| | each respective country patients who have |
| | completed the study without early treatment |
| | discontinuation will be offered to roll over to |
| | M15-997 open label extension (OLE) trial if they |
| | fulfil the in- and exclusion criteria for the M15- |
| | 997 trial. Refer to section 6.2.3. |
| | Next visit and also the last visit after 1st May and |
| | approval of this amendment will be the extended |
| | EOS visit .Termination of trial medication page |
| | should be completed in the eCRF and treatment |
| | completed registered in IRT. |
| Rationale for change | Transition of patients from 1311.13 to M15-997 |
| | study |

| Section to be changed FLOW CHART-extended dosing period Serum pregnancy testing and TB screening add to the EOS visit. Rationale for change Added to the EOS visit because this will be the last visit in the study instead for EOT visit for patients not prematurely discontinued. Section to be changed FLOW CHART-extended dosing period Consent for vital status follow up deleted from EOS visit. Rationale for change No longer applicable as the patients will be | ; |
|---|---|
| to the EOS visit. Rationale for change Added to the EOS visit because this will be the last visit in the study instead for EOT visit for patients not prematurely discontinued. Section to be changed FLOW CHART-extended dosing period Consent for vital status follow up deleted from EOS visit. | ; |
| last visit in the study instead for EOT visit for patients not prematurely discontinued. Section to be changed FLOW CHART-extended dosing period Consent for vital status follow up deleted from EOS visit. | |
| patients not prematurely discontinued. Section to be changed FLOW CHART-extended dosing period Consent for vital status follow up deleted from EOS visit. | |
| Section to be changed FLOW CHART-extended dosing period Description of change Consent for vital status follow up deleted from EOS visit. | |
| Description of change Consent for vital status follow up deleted from EOS visit. | |
| Description of change Consent for vital status follow up deleted from EOS visit. | |
| EOS visit. | |
| Rationale for change No longer applicable as the nation to will be | |
| transferred to the M15-997 and this study will | |
| end. | |
| Section to be changed FLOW CHART-extended dosing period | |
| Description of change •Footnote 4: Variable depending on marketing | |
| approval of BI 655066 deleted | |
| •Footnote 5: If study is ongoing beyond Extend | led |
| visit 18, forthcoming visits should be repeated | |
| cycles as described in Extended visit 6 -18 unti | |
| the patient withdraws, or the end of study is | |
| declared. Visits will be numbered consecutivel | V |
| (Extended visit 19, Extended visit 20,) delet | • |
| | No longer applicable as it is decided when the |
| study will end. | |
| Section to be changed 3.10VERALL TRIAL DESIGN AND PLAN | |
| <b>Description of change</b> Text deleted: The study is planned to continue | ın |
| each country in which it is conducted, until BI | |
| 655066 is approved and available on the market | :t |
| in that country. | ·C |
| Text added: After 01-May-2018 and approval of this protocol amendment in each respective | )1 |
| country, the next study visit will be the Extend | ed |
| EOS visit and therewith the last visit in this stu | |
| Patients who have completed the study without | • |
| early treatment discontinuation will be offered | |
| roll over to M15-997 open label extension (OL | |
| trial if they fulfil the in- and exclusion criteria: | |
| the M15-997 trial. Refer to section 6.2.3. | |
| Rationale for change Transition of patients from 1311.13 to M-15-99 | <del></del> |
| Section to be changed 6.3 End of trial and Extended follow-up period | |
| <b>Description of change</b> Update why and how the 1311.13 study should | Update why and how the 1311.13 study should |
| end | |
| Rationale for change Study drug is not marketed yet and the patient | |

| will be offered to roll over to M15-997 open label |
|----------------------------------------------------|
| extension study and have the opportunity to |
| continue with Risankizumab (BI 655066). |



## APPROVAL / SIGNATURE PAGE

Document Number: c02318676 Technical Version Number: 8.0

**Document Name:** clinical-trial-protocol-version-06

**Title:** An open label extension trial assessing the safety and efficacy of BI 655066/ABBV-066/risankizumab administered subcutaneously in patients with moderate to severe chronic plaque psoriasis.

## Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|---|---|---|
| Approval- | | 30 Jan 2018 14:53 CET |
| Approval- | | 30 Jan 2018 15:50 CET |
| Author- | | 30 Jan 2018 17:39 CET |
| Approval- | | 01 Feb 2018 14:51 CET |
| Verification-Paper Signature<br>Completion | | 01 Feb 2018 15:05 CET |

Boehringer IngelheimPage 2 of 2Document Number: c02318676Technical Version Number:8.0

(Continued) Signatures (obtained electronically)

| Meaning of Signature | Signed by | Date Signed |
|----------------------|-----------|-------------|
|----------------------|-----------|-------------|